#### **RTOG 1205**

# RANDOMIZED PHASE II TRIAL OF CONCURRENT BEVACIZUMAB AND RE-IRRADIATION VERSUS BEVACIZUMAB ALONE AS TREATMENT FOR RECURRENT GLIOBLASTOMA

This trial is part of the National Clinical Trials Network (NCTN) program, which is sponsored by the National Cancer Institute (NCI). The trial will be led by NRG Oncology with the participation of the network of NCTN organizations: the Alliance for Clinical Trials in Oncology; ECOG-ACRIN Medical Group; and SWOG.

**Study Chairs** (8/24/15)

## Principal Investigator/Radiation Oncology

Christina Tsien, MD Department of Radiation Oncology Washington University in St. Louis 4921 Parkview Place, Campus Box 8224

St. Louis, MO 63110

Phone: 314-362-8567/Fax: 314-362-8521

Email: <a href="mailto:ctsien@radonc.wustl.edu">ctsien@radonc.wustl.edu</a>

Medical Oncology Co-Chair

Jeffrey Raizer, MD Northwestern University 710 N. Lake Shore Drive Abbott Hall, Room 1123 Chicago, IL 60611

Phone: 312-503-4724/Fax: 312-908-5073

E-mail: Jraizer@nm.org

Senior Statistician
Peixin Zhang, PhD
NRG Oncology
1818 Market Street, Suite 1720

Philadelphia, PA 19103

Phone: 215-940-8881/Fax: 215-928-0153 Email: ZhangP@NRGOncology.org Radiation Oncology Co-Chair

Adam P. Dicker, MD, PhD Department of Radiation Oncology Jefferson Medical College of Thomas Jefferson University

111 South 11th Street Philadelphia, PA 19107-5097

Phone: 215-955-6700/Fax: 215-503-0013

E-mail: adam.dicker@jefferson.edu

Medical Physics Co-Chair Martha M. Matuszak, PhD University of Michigan 1500 E. Medical Center Drive

Ann Arbor, MI 48109

Phone: 734-936-4309/Fax: 734-936-7859 E-mail: marthamm@med.umich.edu

#### **Document History**

| | Version/Update Date | Broadcast Date |
|------------------|---------------------|--------------------|
| Amendment 8 | October 3, 2016 | October 17, 2016 |
| Closure | | |
| Amendment 7 | September 3, 2015 | April 28, 2016 |
| Amendment 7 | September 3, 2015 | September 21, 2015 |
| Amendment 6 | August 24, 2015 | September 21, 2015 |
| Amendment 5 | October 9, 2014 | November 3, 2014 |
| Amendment 4 | June 23, 2014 | November 3, 2014 |
| Amendment 3 | April 15, 2014 | May 1, 2014 |
| Amendment 2 | February 27, 2014 | May 1, 2014 |
| Amendment 1 | November 20, 2013 | December 4, 2013 |
| Activation | October 10, 2012 | December 20, 2012 |
| Group Activation | October 10, 2012 | November 5, 2012 |

Protocol Agents (11/20/13)

| Agent | Supply | NSC# | IND# |
|-------------|------------|------|--------|
| Bevacizumab | Commercial | N/A | Exempt |

| Participating Sites (11/20/13) |
|---|
| US Only |
| ☐ Canada Only |
| US and Canada □ □ |
| Approved International Member Sites |

NRG Oncology 1-800-227-5463, ext. 4189

This protocol was designed and developed by NRG Oncology. It is intended to be used only in conjunction with institution-specific IRB approval for study entry. No other use or reproduction is authorized by NRG Oncology nor does NRG Oncology assume any responsibility for unauthorized use of this protocol.

(10/3/16)

| CTSU CONTACT INFORMATION | | |
|---|---|---|
| For regulatory requirements: | For patient enrollments: | For study data submission: |
| Regulatory documentation can | Please refer to the patient | See Protocol Section 12.0 for |
| be submitted to the CTSU via: | enrollment section of the protocol | data submission |
| | for instructions on using the | |
| ONLINE: | Oncology Patient Enrollment | Do <u>not</u> submit study data or |
| Regulatory Submission Portal | Network (OPEN) which can be | forms to CTSU Data Operations. |
| (Sign in at <u>www.ctsu.org</u> , | accessed at | Do not copy the CTSU on data |
| and select the Regulatory | https://www.ctsu.org/OPEN_SYS | submissions. |
| Submission sub-tab under the | TEM/ or https://OPEN.ctsu.org. | |
| Regulatory tab.) | 0 1 1 1 0 0 0 0 1 | |
| EMAIL: | Contact the CTSU Help Desk | |
| CTSURegulatory@ctsu.coccg. | with any OPEN-related questions | |
| org (regulatory documentation | at <a href="mailto:ctsucontact@westat.com">ctsucontact@westat.com</a> | |
| only)<br><b>FAX</b> : | | |
| 215-569-0206 | | |
| MAIL: | | |
| CTSU Regulatory Office | | |
| 1818 Market Street, Suite 1100 | | |
| Philadelphia, PA 19103 | | |
| 1 1 madelpina, 1 7 10 100 | | |
| For regulatory questions call | | |
| the CTSU Regulatory Help | | |
| Desk at 1-866-651-CTSU | | |

The most current version of the **study protocol and all supporting documents** must be downloaded from the protocol-specific Web page of the CTSU Member Web site located at <a href="https://www.ctsu.org">https://www.ctsu.org</a>. Access to the CTSU members' website is managed through the Cancer Therapy and Evaluation Program - Identity and Access Management (CTEP-IAM) registration system and requires user log on with CTEP-IAM username and password.

For clinical questions (i.e. patient eligibility or treatment-related): Contact the Study PI of the Lead Protocol Organization.

- For non-clinical questions (i.e. unrelated to patient eligibility, treatment, or clinical data submission) contact the CTSU Help Desk by phone or e-mail:
- CTSU General Information Line 1-888-823-5923, or <a href="mailto:ctsucontact@westat.com">ctsucontact@westat.com</a>. All calls and correspondence will be triaged to the appropriate CTSU representative.

The CTSU Website is located at https://www.ctsu.org.

## TABLE OF CONTENTS

| | MABILITY CHECKLIST | |
|---|---|---|
| | INTRODUCTION | |
| 1.0 | | |
| 1.1<br>1.2 | OverviewSafety, Efficacy, and Rationale for Combination of Bevacizumab and Re-Irradiation | |
| 1.2 | Salety, Efficacy, and Rationale for Combination of Bevacizumab and Re-irradiation | 14 |
| 2.0 | OBJECTIVES | |
| 2.1 | Primary Objective | |
| 2.2 | Secondary Objectives | 15 |
| 3.0 | PATIENT SELECTION | |
| 3.1 | Conditions for Patient Eligibility | |
| 3.2 | Conditions for Patient Ineligibility | 17 |
| 4.0 | PRETREATMENT EVALUATIONS/MANAGEMENT | |
| 4.1 | Highly Recommended Evaluations | 17 |
| 5.0 | REGISTRATION PROCEDURES | 18 |
| 5.1 | Pre-Registration Requirements for Image-Guided Radiotherapy (IGRT) Treatment Approach) | |
| 5.2 | Pre-Registration Requirements for IMRT Treatment Approach | |
| 5.3 | Pre-Registration Requirements for 3D-CRT Treatment Approach | |
| 5.4 | Pre-Registration Requirements for Proton Treatment Approach | |
| 5.5<br>5.6 | Digital RT Data Submission Using TRIAD | |
| 5.7 | Regulatory Pre-Registration Requirements | |
| 0.0 | DADIATION THEDADY | 01 |
| 6.0<br>6.1 | RADIATION THERAPY | |
| 6.2 | Technical Factors [Equipment, energies] | |
| 6.3 | Localization, Simulation, and Immobilization | |
| 6.4 | Treatment Planning/Target Volumes | |
| 6.5 | Critical Structures | |
| 6.6 | Documentation Requirements | |
| 6.7 | Compliance Criteria | |
| 6.8 | R.T. Quality Assurance Reviews | |
| 6.9 | Radiation Therapy Adverse Events | |
| 6.10 | Radiation Therapy Adverse Event Reporting | |
| 7.0 | DRUG THERAPY | 26 |
| 7.1 | Treatment | |
| 7.2 | Bevacizumab Agent Information | |
| 7.3 | Bevacizumab Dose Modifications | |
| 7.4 | Modality Review | 35 |
| 7.5 | Adverse Events | |
| 7.6 | CTEP-AERS Expedited Reporting Requirements | 37 |
| 8.0 | SURGERY | 39 |
| 9.0 | OTHER THERAPY | 39 |
| 9.1 | Permitted Supportive Therapy | |

| 9.2 | Non-permitted Supportive Therapy | 39 |
|------|------------------------------------------------------------|----|
| 10.0 | TISSUE/SPECIMEN SUBMISSION | 39 |
| 10.1 | Tissue/Specimen Submission | |
| 10.2 | Specimen Collection for Banking and Translational Research | 39 |
| 10.3 | Reimbursement | |
| 10.4 | Confidentiality/Storage | |
| 11.0 | PATIENT ASSESSMENTS | 42 |
| 11.1 | Study Parameters | |
| 11.2 | Measurement of Response | |
| 11.3 | Criteria for Evaluation of Therapy Effectiveness | 43 |
| 11.4 | RANO Response Criteria | |
| 11.5 | Criteria for Discontinuation of Protocol Treatment | |
| 12.0 | DATA COLLECTION | 46 |
| 12.1 | Summary of Data Submission | |
| 12.2 | Summary of Dosimetry Digital Data Submission | |
| 13.0 | STATISTICAL CONSIDERATIONS | 47 |
| 13.1 | Study Endpoints | |
| 13.2 | Sample Size and Power Justification | |
| 13.3 | Patient Accrual | |
| 13.4 | Patient Stratification and Randomization | 48 |
| 13.5 | Analyses Plans | 48 |
| 13.6 | Gender and Minorities | |
| REFE | RENCES | 51 |
| | NDIX I | |
| | NDIX II | |
| | NDIX III | |

## **NRG ONCOLOGY**

## **RTOG 1205**

## Randomized Phase II Trial of Concurrent Bevacizumab and Re-Irradiation Versus Bevacizumab Alone as Treatment for Recurrent Glioblastoma

## **SCHEMA** (4/15/14)

#### **Bevacizumab-Naïve Recurrent GBM Patients:**

| Age 1. <50 2. ≥50 R Karnofsky performance status 1. 60 2. 70-80 3. 90-100 Recent resection 1.Yes 2. No/biopsy only R R A A N Arm 1: Bevacizumab alone q 2 weeks (control arm) Arm 2: Hypofractionated radiotherapy 35 Gy in 10 fractions with concurrent Bevacizumab q 2 weeks (experimental arm) |
|---|
|---|

See  $\underline{\text{Section 5.0}}$  for radiation therapy credentialing requirements. See  $\underline{\text{Section 7.0}}$  for details/doses of bevacizumab.

<u>Patient Population</u>: (See <u>Section 3.0</u> for Eligibility)

Patients with recurrent glioblastoma or variant (gliosarcoma or giant cell glioblastoma etc).

**Required Sample Size: 178** 

## ELIGIBILITY CHECKLIST (10/9/14) 

## NRG Oncology Institution # RTOG 1205 Case #

| (Y) | 1. | Does the patient have histologically proven diagnosis of glioblastoma or variants per <u>section 3.1.1</u> ? |
|---|---|---|
| (Y/NA) | 2. | Does patient have progression on contrast-enhanced MRI/CT within 21 days prior to registration as defined in <u>section 3.1.1</u> , bullet 1? |
| (Y/N) | 3. | Is there an interval of 6 months or greater between completion of prior radiotherapy and registration? (Y) If No, was one or more of the criteria in section 3.1.1 a, b or c met? |
| (Y/N) | 4. | Does the patient have a prior history of standard dose CNS radiation as defined in section 3.1.2? (Y) If No, was one or more of the criteria in section 3.1.1 a, b or c met? |
| (Y/NA) | 5. | Has patient recovered from the toxic effects of prior therapy? |
| (Y/NA) | 6. | If patient received prior investigational agent(s) and/or prior cytotoxic therapy was there a minimum time of 28 days prior to registration? With the exceptions of vincristine (minimum time of 14 days), nitrosoureas (minimum time of 42 days) and procarbazine (minimum time of 21 days) |
| (Y/N) | 7. | Did the patient have a recent resection (within 5 weeks prior to registration) of the glioblastoma? If Y: (Y) Has the patient recovered from the effects of surgery? (Y/NA) Has a minimum of 7 days elapsed for core or needle biopsy? (Y) Was a postoperative or intraoperative scan performed prior to registration? |
| (Y) | 8. | Was a history and physical examination completed within 14 days prior to registration? |
| (Y) | 9. | Is the Karnofsky performance status greater than or equal to 60 within 14 days prior to registration? |
| (Y) | 10. | Is the patient's age ≥18? |
| (Y) | 11. | Was a CBC with differential obtained within 14 days prior to registration with adequate bone marrow function as defined in <a href="mailto:section3.1.8">section 3.1.8</a> ? |
| (Y) | 12. | Is there adequate liver and renal function within 14 days prior to registration as defined in <a href="mailto:section3.1.8">section 3.1.8</a> ? |
| (N) | 13. | Does the patient have proteinuria within 14 days of registration as defined in section 3.1.9? |
| (N/NA) | 14. | Is the patient pregnant or nursing? |

## ELIGIBILITY CHECKLIST (9/3/15) 

## NRG Oncology Institution # RTOG 1205 Case #

| (Y/NA) | 15. Was a pregnancy test done within 7 days before registration? |
|---|---|
| (Y/NA) | 16. Is the patient willing to practice effective contraception while on study treatment<br>and 6 months after? (women of childbearing potential and men) |
| (Y/N) | 17. Is the patient on full dose anticoagulants? If Y: |
| | (N) Does the patient have active bleeding or a pathological condition that carries a high risk of bleeding? (Y) Is there an in-range INR (usually between 2 and 3) on a stable dose of oral anticoagulant or on a stable dose of low molecular weight heparin within 14 days prior to registration? |
| (Y) | 18. Did the patient provide study-specific informed consent prior to study entry? |
| (N) | 19. Has the patient had more than 3 relapses? |
| (N) | 20. Is there infratentorial or leptomeningeal evidence of recurrent disease? |
| (N) | 21. Does the patient have a recurrent or persistent tumor greater than 6 cm in maximum diameter? |
| (N) | 22. Has the patient had prior therapy with an inhibitor of VEGF or VEGFR (including bevacizumab)? |
| (Y/N) | 23. Has the patient had prior invasive malignancy (except non- melanomatous skin cancer)? If Y: |
| | (Y) Has the patient been disease free for a minimum of 1 year |
| (N) | 24. Does the patient have severe active co-morbidity as in defined in <u>3.2.6</u> .? |
| (N) | 25. Does the patient have prior allergic reaction to the study drug (Bevacizumab)? |
| (N) | 26. Does the patient have prior history of hypertensive crisis or hypertensive encephalopathy? |
| (N) | 27. Does the patient have a history of a non-healing wound, ulcer or bone fracture within 90 days (3 months) prior to registration? |
| (N) | 28. Has the patient had gastrointestinal bleeding or any other hemorrhage/bleeding event CTCAE, v.4 grade 3 or greater within 30 days prior to registration? |
| (N) | 29. Has the patient had major surgical procedure, open biopsy or significant<br>traumatic injury within 28 days prior to registration (with the exception of<br>craniotomy)? |

## ELIGIBILITY CHECKLIST (11/5/12) 

NRG Oncology Institution # RTOG 1205 Case #

\_\_\_\_(Y/N) 20.

(Y/N) 21.

The following questions will be asked at Study Registration: IMRT CREDENTIALING AND IGRT CREDENTIALING (for reduced margins only) IS REQUIRED BEFORE REGISTRATION. PROTON CREDENTIALING IS REQUIRED IF USING PROTONS. 1. Institutional person randomizing case. (Y) 2. Has the Eligibility Checklist been completed? \_\_\_\_(Y) 3. In the opinion of the investigator, is the patient eligible? 4. Date informed consent signed 5. Patient Initials (First Middle Last) 6. Verifying Physician 7. Patient ID Date of Birth 8. 9. Race 10. Ethnicity 11. Gender 12. Country of Residence 13. Zip Code (U.S. Residents) 14. Method of Payment Any care at VA or Military Hospital? 15. 16. Calendar Base Date 17. Randomization date 18. Medical oncologist's name (Y/N) 19. Have you obtained the patient's consent for his or her tissue to be kept for use in research to learn about, prevent, treat, or cure cancer?

research to learn about, prevent, treat, or cure cancer?

research to learn about, prevent, treat, or cure cancer?

Have you obtained the patient's consent for his or her blood to be kept for use in

Have you obtained the patient's consent for his or her urine to be kept for use in

## ELIGIBILITY CHECKLIST (11/5/12) 

NRG Oncology Institution # RTOG 1205 Case #

| (Y/N) | 22. | Have you obtained the patient's consent for his or her tissue to be kept for use in research about other health problems (for example: causes of diabetes, Alzheimer's disease, and heart disease)? |
|---|---|---|
| (Y/N) | 23. | Have you obtained the patient's consent for his or her blood to be kept for use in research about other health problems (for example: diabetes, Alzheimer's disease, or heart disease). |
| (Y/N) | 24. | Have you obtained the patient's consent for his or her urine to be kept for use in research about other health problems (for example: causes of diabetes, Alzheimer's disease, and heart disease)? |
| (Y/N) | 25. | Have you obtained the patient's consent to allow someone from this institution to contact him or her in the future to take part in more research? |
| | 26. | Patient's age (<50/≥50):<br>(1) <50<br>(2) ≥50 |
| | 27. | Karnofsky performance status:<br>(1) 70-80<br>(2) 90-100<br>(3) 60 |
| | 28. | (Y/N-biopsy only): Recent resection |
| (Y/N) | 29. | Did the patient participate in a previous RTOG GBM trial that collected MGMT methylation status? If yes, what was the RTOG study number? If yes, what was the patient ID number on the RTOG trial mentioned above? |
| (Y/N) | 30. | Did the patient have MGMT analysis performed as routine care by a treating physician outside of an RTOG GBM trial (or that was collected during an RTOG trial but <b>not required</b> per protocol)? If yes, what was the result of MGMT analysis? (1) Methylated (2) Unmethylated (3) Invalid |
| (Y/N) | 31. | Will IGRT be used for patient positioning? |
| (Y/N) | 32. | Will IGRT be used for patient positioning and margin reduction? |
| | 33. | Specify treatment techniques/machine: (1) 3D-CRT (2) IMRT (3) Cyberknife (4) Protons |

## ELIGIBILITY CHECKLIST (11/5/12) 

NRG Oncology Institution # RTOG 1205 Case #

| The Eligibility Checklist must be completed in its entirety | prior to web registration. The completed, signed, |
|---|---|
| and dated checklist used at study entry must be retained | in the patient's study file and will be evaluated |
| during an institutional NCI/NRG Oncology audit. | |
| - | |
| Completed by | Date |
| | <u> </u> |

#### 1.0 INTRODUCTION

#### 1.1 Overview

Glioblastoma is the most common lethal primary brain tumor in adults (Brandes 2003). Despite optimal treatment including surgery, chemotherapy, and radiation, median survival of patients with glioblastoma is 14 months. The majority of patients will develop recurrence at a median of 8 months post treatment (Stupp 2005).

Patients with recurrent glioblastoma have poor prognoses and have been treated with various modalities including resection, chemotherapy, or re-irradiation. Prior phase II chemotherapy trials were associated with a 6-month progression-free survival of 15% and a median survival of 25 weeks (Wong 1999, Carson 2007). In 2009, bevacizumab, a humanized monoclonal antibody which targets VEGF, was approved by the FDA as a single agent for recurrent glioblastoma.

Vascular proliferation is a notable feature in glioblastoma; therefore, targeting the vascular endothelial growth factor (VEGF) is a logical treatment approach (Jain 2007). Anti-VEGF therapy can inhibit new vessel growth, lead to vascular regression and vascular normalization, as well as directly affect tumor cell function (Ellis 2008). Antiangiogenic therapies rapidly normalize leaky abnormal tumor vessels and therefore decrease vasogenic edema as well as the patient's dependence on corticosteroids. This effect may lead to significant improvement in the patient's quality of life (Vredenburgh 2010).

Several clinical trials have evaluated the safety and efficacy of bevacizumab alone or in combination with chemotherapy in recurrent gliomas. A single-institution phase II trial demonstrated increased response rates and prolonged 6-month progression-free survival (Vredenburgh 2007a; Vredenburgh 2007b). Thirty-two patients with recurrent grade III-IV glioma (Vredenburgh 2007a) received bevacizumab and irinotecan, showing promising activity with a 6-month progression-free survival of 38%. The median overall survival limited to grade IV patients was 9.2 months.

In a phase II trial, 48 heavily pretreated recurrent glioblastoma patients received single-agent bevacizumab, with a median progression-free survival of 16 weeks, 6-month progression-free survival of 29%, and a response rate of 35% based on Macdonald criteria (Kreisl 2009). A subsequent randomized, non-comparative phase II trial (BRAIN study) was performed and led to the FDA approval of single-agent bevacizumab. Patients with recurrent glioblastoma in first or second relapse were randomized to either bevacizumab 10 mg/kg every 2 weeks alone (85 patients) or in combination with irinotecan (82 patients). The estimated 6-month progression-free survival rate was 42.6% and 50.3%, respectively. Median overall survival was 9.2 and 8.7 months, respectively. The majority of patients in this trial had partial or complete resection (91.8% and 91.5%, respectively). A minority of patients (8% and 13%, respectively) were enrolled ≤3 months following radiotherapy, while 20% and 10%, respectively, were enrolled ≤3 months following surgery. Overall, treatment was well tolerated; adverse events related to bevacizumab included hypertension, fatique, and deep vein thrombosis. There was no clear increase in efficacy with the addition of irinotecan; however, there was increased toxicity (Friedman 2009). Despite the significant increase in response rates and 6-month progression-free survival with single-agent bevacizumab, the median overall survival remains 8 to 9 months.

Several phase II trials have attempted to combine bevacizumab with other chemotherapy agents, with no significant improvement in outcome. These agents include daily low-dose temozolomide, etoposide, erlotinib, and nitrosourea. In fact, these trials identified increased toxicity with no improvement in efficacy (Verhoeff 2010; Gilbert 2009; Hasselbach 2010; Reardon 2009; Sathornsumetee 2010). Response rates to chemotherapy following bevacizumab failure are exceptionally poor. Salvage chemotherapy provided only transient tumor control with an estimated 6-month progression-free survival of 2% (Quant 2009). Enrollment in a clinical trial for patients with recurrent glioblastoma should be the standard clinical practice and highlights the pressing need to identify novel strategies.

Salvage re-irradiation has long been offered as a treatment modality (Hudes 1999, Kim 1997, Laing 1993, Grosu 2005, Lederman 2000). Prior results obtained from over 300 glioblastoma patients confirmed a 6-month progression-free survival ranging from 28% to 39% and a median 1-year overall survival of 26% ranging from 18% to 46% (Combs 2005, Nieder 2008, Fogh 2010). However, recent advances in RT techniques including fractionated stereotactic radiotherapy (FSRT), protons, and IMRT, now allow for highly conformal treatment, which has the potential to significantly reduce the toxicity associated with re-irradiation (Fogh 2010).

Several studies report an improvement in 6-month functional status as well as a reduction and discontinuation of corticosteroid usage (Laing 1993; Kim 1997; Nieder 2008; VanderSpek 2008). Late CNS toxicity was uncommon especially following FSRT. Combs et al reported on 172 recurrent gliomas with a median time from RT to re-radiation of 10 months. Median tumor size for glioblastoma tumors was 47.7 cc. RT dose was 36 Gy in 2 Gy fractions given 5 fractions per week. Progression-free survival for 59 glioblastoma patients following re-irradiation was 5 months, with a median overall survival of 8 months. Factors associated with improved outcome included histology, extent of initial resection, and age at primary diagnosis. Treatment was well tolerated, with 1 incidence of radiation necrosis (Combs 2005).

Fogh et al reported on 147 high-grade glioma patients treated with FSRT delivering 35 Gy in 10 fractions. Median time to re-irradiation was 8 months. Somewhat surprisingly, and in contrast with other reports, patients who received irradiation within 6 months of initial diagnosis did not demonstrate an inferior survival. Median tumor volume was 22 cc. Eighty-four patients underwent salvage surgery prior to re-irradiation. Forty-eight patients received concurrent chemotherapy such as temozolomide. Median survival was 11 months. Treatment was well tolerated. Multivariate analysis suggested younger age and smaller tumor volumes were associated with improved outcome (Fogh 2010).

There is a clear rationale for combining bevacizumab with re-irradiation to increase the therapeutic ratio through increased antitumor and antivascular effects (Provencio 2010; Lee 2000). Preclinical data suggest that VEGF is up-regulated in response to radiation; therefore, the use of antiangiogenic agents combined with radiation may sensitize both tumors and associated vasculature to RT (Gorski 1999). Preclinical studies have demonstrated that antiangiogenic agents may uniquely target the radio-resistant and highly tumorigenic cancer stem cells by disrupting vascular niches harboring cancer stem cells (Hovinga 2010). Due to its potential radioprotective effects, especially the phenomenon of vascular stabilization, the addition of bevacizumab may also reduce the toxicity associated with re-irradiation by reducing risk of radiation necrosis (Levin 2011). Several phase II and phase III trials have reported on the initial safety and tolerability of combining bevacizumab and temozolomide with radiotherapy in primary glioblastoma patients (Lai 2010; Vredenburgh 2011).

Preliminary evidence suggests improved outcome with the addition of concurrent and adjuvant bevacizumab to re-irradiation. Gutin et al published results regarding 25 patients with recurrent grade III-IV gliomas using FSRT and concurrent bevacizumab; with a reported 6-month progression-free survival of 65% and median overall survival of 12.5 months. Median time to radiation was 15 months. Enhancing tumor volume was ≤ 3.5 cm in maximum diameter. Treatment was well tolerated. There was no incidence of radiation necrosis and no additional need for corticosteroids following radiation (Gutin 2009).

The Duke group recently reported its single-institution retrospective data on 63 patients with recurrent high-grade gliomas, including 49 glioblastoma patients treated with re-irradiation using SRS techniques combined with bevacizumab therapy. The treatment regimen was noted to be well tolerated. Median time to re-irradiation was 19.6 months. Mean number of systemic therapies prior to SRS was 3.6 and mean number of therapies following SRS was 2.9. Median target volume was 4.8 cc. The 1-year overall survival in glioblastoma patients who received adjuvant (concurrent with or after SRS) bevacizumab was 50% vs. 22% for patients not receiving adjuvant

bevacizumab (p= 0.005). Both age < 50 years and performance status > 70 were associated with improved overall survival (Cuneo 2011).

Retrospective single-institutional experience in high-grade glioma patients treated with FSRT using 36 Gy in 18 fractions, with concurrent bevacizumab, followed by maintenance bevacizumab was recently reported. Overall survival appeared better in patients receiving bevacizumab (12.1 months) than those who had received either re-irradiation alone or concurrent with temozolomide (8.0 months). Treatment was well tolerated, with no incidence of radiation necrosis and one incidence of wound dehiscence (Niyazi 2010).

Based on the long history and clinical experience of re-irradiation of recurrent glioblastoma, we wish to obtain prospective multi-institutional safety and efficacy data regarding the combination of bevacizumab and re-irradiation in improving overall survival in bevacizumab-naïve recurrent glioblastoma patients.

Therefore, the primary aim of this study is to provide preliminary evidence of an overall survival benefit with the addition of re-irradiation in combination with bevacizumab for patients with recurrent glioblastoma in a multi-institutional setting, in the context of a phase II randomized trial that will require further confirmation in a phase III trial.

#### **1.1.1** Significance of the Current Study

RTOG 1205 is important in potentially changing the paradigm of treatment in recurrent glioblastoma. Despite numerous randomized chemotherapy studies as well as novel targeted agents studied to date, no regimens have shown significant improvement in overall survival compared to bevacizumab alone. Single-agent bevacizumab is currently the mainstay of treatment in recurrent glioblastoma, but the overall survival remains limited at approximately 8 to 9 months. Responses to therapy following bevacizumab failures are extremely poor. Preclinical data suggest that a resistant and invasive phenotype develops following bevacizumab failure, and salvage therapy remains ineffective in this context; therefore, this latter patient group will NOT be included in our trial.

The goal of this study is to test the hypothesis that re-irradiation combined with an effective targeted agent, bevacizumab, will improve the overall survival of bevacizumab-naïve recurrent glioblastoma patients. This trial will also be the first prospective multi-institutional study to evaluate survival, response, and patterns of failure following re-irradiation. Further, if this trial is positive, the implication is that higher radiotherapy doses are potentially feasible and safe, and therefore, the addition of bevacizumab and re-irradiation in recurrent gliomas may provide the preliminary proof of principle to further study dose-escalated radiation in combination with bevacizumab in the upfront treatment of glioblastoma. Additionally, this trial could also potentially set the stage for testing additional chemotherapeutic and/or targeted agents with radiation in the recurrent glioblastoma setting. This could provide preliminary clinical data to move promising agents in the upfront setting in a more efficient manner.

#### 1.2 Safety, Efficacy, and Rationale for Combination of Bevacizumab and Re-Irradiation

The safety and efficacy of hypofractionated stereotactic irradiation in combination with bevacizumab for recurrent glioblastoma was reported by Gutin et al (2009). The results were promising, with a 6-month progression-free survival of 65% and a median overall survival of 12.5 months. There were no incidences of radiation necrosis noted and there was no need for additional corticosteroids following treatment. The treatment was also safe and well tolerated. Grade 3 toxicity, including intratumor hemorrhage, wound dehiscence, and bowel perforation, was noted in 12% of patients. Retrospective results of hypofractionated stereotactic radiation alone using 35 Gy in 10 fractions in 147 high-grade glioma patients were reported by Fogh et al (2010). Median survival was 11 months. This underscores the safety and tolerability of this approach.

RTOG 0625, a phase II randomized study of bevacizumab and irinotecan or temozolomide, enrolled 123 patients and was recently published in abstract form (Gilbert 2009). ACRIN 6637

provided central review of all pre-treatment MRIs. Analysis of the pre-treatment MRI confirmed that over 90% of cases had an initial post-contrast T1 MRI tumor diameter of 5 cm or less. A statistical analysis was performed using this inclusion criteria (limiting to 5 cm or less), and demonstrated a median overall survival of 9.4 months for patients receiving bevacizumab and temozolomide and 7.6 months for patients receiving bevacizumab and irinotecan (Wang, RTOG 0625 summary analysis unpublished data). This preliminary analysis confirms the median survival of recurrent glioblastoma treated with bevacizumab at approximately 9 months and a basis for the inclusion of tumors limited in size to 5 cm diameter.

Re-irradiation using the newer SRS techniques delivers higher doses of irradiation to a considerably more precise target volume, in a single fraction, and with a steep dose gradient beyond the tumor. In several series reporting on these novel SRS techniques, overall survival was 9 to 11 months. Because of the potential CNS toxicity associated with a single-fraction treatment or treatment with very few fractions of large dose per fraction, patients selected for this therapy must have small, limited volume recurrences. Fractionation leads to improvement of the therapeutic ratio by reducing the risk to normal tissues compared with single-fraction treatments, especially for larger tumors (3 to 5 cm) (Brenner 1997, Cho 1999). The linear quadratic (LQ) model has been used to calculate the biological equivalent dose using a tumor alpha/beta ratio of 10 Gy (Mayer 2008). The effect on late normal tissue was calculated using an alpha/beta ratio of 3 Gy. The proposed schema in this study of 35 Gy in 10 fractions was directly compared to the 30 Gy in 5 fractions used by Gutin et al and was predicted using biologic modeling to have similar antitumor efficacy (47.2 versus 48 Gy with alpha-beta of 10 Gy). However, the 35 Gy in 10 fractionation scheme is much more favorable in regards to risk of late normal tissue toxicity and is likely better tolerated for larger tumors.

#### 2.0 OBJECTIVES

## 2.1 Primary Objective

To establish an improvement in overall survival in recurrent GBM patients receiving bevacizumab and re-irradiation compared with patients receiving bevacizumab alone.

## 2.2 Secondary Objectives

- **2.2.1** To estimate and compare the rate of objective response in patients with measurable disease.
- **2.2.2** To estimate and compare the 6-month progression-free survival rate.
- **2.2.3** To estimate and compare progression-free survival.
- **2.2.4** To estimate and compare the rate of treatment adverse events.
- 2.2.5 To estimate and compare the rate of ≥grade 3 acute or delayed CNS toxicity.

#### 3.0 PATIENT SELECTION

#### NOTE: PER NCI GUIDELINES, EXCEPTIONS TO ELIGIBILITY ARE NOT PERMITTED

#### 3.1 Conditions for Patient Eligibility (8/24/15)

For questions concerning eligibility, please contact the study data manager.

- **3.1.1** Histopathologically proven diagnosis of glioblastoma or variants (gliosarcoma, giant cell glioblastoma etc). Patients will be eligible if the original histology was lower-grade glioma and a subsequent diagnosis of glioblastoma or gliosarcoma is made.
  - Patients who did not have recent surgery for their glioblastoma must have shown unequivocal radiographic evidence for tumor progression by contrast-enhanced MRI scan (or CT scan for patients with non-compatible devices) within 21 days prior to registration as defined in Section 11.4.1.

Note: Patients who did have surgery with a post-operative contrast-enhanced scan falling outside the 5-week window prior to registration, per definition of recent surgery in 3.1.4, must have a repeat MRI scan (or CT scan for patients with non-compatible devices) within 21 days prior to registration.

• Patients must have passed an interval of 6 months or greater between <u>completion</u> of prior radiotherapy and registration. If patients have not passed an interval of at least 6 months, they may still be eligible if they meet one or more of the following criteria:

- a) New areas of tumor outside the original radiotherapy fields as determined by the investigator, or
- b) Histologic confirmation of tumor through biopsy or resection, or
- c) Nuclear medicine imaging, MR spectroscopy, or MR perfusion imaging consistent with true progressive disease, rather than radiation necrosis obtained within 28 days of registration AND an interval of at least 90 days between completion of radiotherapy and registration.
- Patients unable to undergo MR imaging because of non-compatible devices can be enrolled provided CT scans are obtained and are of sufficient quality. Patients without non-compatible devices may not use CT scans performed to meet this requirement.
- **3.1.2** Prior history of standard dose CNS radiation of 60 Gy in 30 fractions or 59.4 Gy in 1.8 Gy fractions, or equivalent or lower doses.
  - Patients who have received prior treatment with non-standard RT dose and fractionation, interstitial brachytherapy, stereotactic radiosurgery, etc. are eligible as long as the criterion in 3.1.1 a, b, or c is met or approved by principal investigator.
- **3.1.3** Patients must have recovered from the toxic effects of prior therapy, and there must be a minimum time of 28 days prior to registration from the administration of any investigational agent or prior cytotoxic therapy with the following exceptions:
  - 14 days from administration of vincristine
  - 42 days from administration of nitrosoureas
  - 21 days from administration of procarbazine
- **3.1.4** Patients having undergone recent resection of their glioblastoma (within 5 weeks prior to registration) must have recovered from the effects of surgery. For CNS related core or needle biopsies, a minimum of 7 days must have elapsed prior to registration.

Residual disease following resection of recurrent glioblastoma is not mandated for eligibility into the study. To best assess the extent of residual disease post-operatively, a post-operative or intra-operative MRI scan (or CT scan for patients with non-compatible devices) must be performed prior to registration and should be within 96 hours post surgery (although 24 hours would be optimum).

- **3.1.5** History/physical examination, including neurologic examination, within 14 days prior to registration
- **3.1.6** Karnofsky performance status ≥ 60 within 14 days prior to registration
- **3.1.7** Age ≥ 18
- **3.1.8** CBC/differential obtained within 14 days prior to registration, with adequate bone marrow function. Adequate bone marrow reserve as follows:
  - Absolute neutrophil count (ANC) ≥ 1,500 cells/mm<sup>3</sup>
  - Platelets ≥ 75.000 cells/mm<sup>3</sup>
  - Hemoglobin ≥ 9.0 g/dl (Note: The use of transfusion or other intervention to achieve Hgb ≥ 9.0 g/dl is acceptable.)
- **3.1.9** Acceptable liver (total bilirubin  $\leq$  2.0 mg/dL, and SGOT or AST  $\leq$  2.5 times the upper limit of normal) and renal function (serum creatinine  $\leq$  1.8 mg/dL) within 14 days prior to registration.
  - Urine protein: creatinine (UPC) ratio < 1.0 within 14 days prior to registration <u>OR</u> urine dipstick for proteinuria ≤ 2+ (patients discovered to have > 2+ proteinuria on dipstick urinalysis at baseline must have a UPC ratio done that is <1.0 to be eligible. If the UPC ratio is ≥ 1.0 then the patients should undergo a 24-hour urine collection and must demonstrate ≤ 1g of protein in 24 hours to be eligible).

| Note: UPC ratio of | spot urine is an estimation of the 24-hour urine protein excretion; a UPC |
|---|---|
| ratio of 1 | is roughly equivalent to a 24-hour urine protein of 1 gm. UPC ratio is |
| calculated | using one of the following formulas: |
| | [urine protein]/[urine creatinine]: if both protein and creatinine are |
| | reported in mg/dL |
| | [(urine protein) x0.088]/[urine creatinine]: if urine creatinine is reported in |
| | mmol/L |

- **3.1.10** Patients must not be pregnant (positive pregnancy test) or breast feeding; pregnancy test must be done within 7 days prior to registration. Effective contraception (men and women) must be used in patients of child-bearing potential while on study treatment and for 6 months after.
- **3.1.11** Patients on full-dose anticoagulants (e.g., warfarin or LMW heparin) must meet both of the following criteria:
  - No active bleeding or pathological condition that carries a high risk of bleeding (e.g., tumor involving major vessels or known varices)
  - In-range INR (usually between 2 and 3) on a stable dose of oral anticoagulant or on a stable dose of low molecular weight heparin, within 14 days prior to registration
- **3.1.12** Patient must be able to provide study-specific informed consent prior to study entry.

#### 3.2 Conditions for Patient Ineligibility (4/15/14)

- **3.2.1** More than three relapses
- **3.2.2** Infratentorial, or leptomeningeal evidence of recurrent disease
- **3.2.3** Recurrent or persistent tumor greater than 6 cm in maximum diameter
- **3.2.4** Prior therapy with an inhibitor of VEGF or VEGFR (including bevacizumab)
- **3.2.5** Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 1 year (for example, carcinoma *in situ* of the breast, oral cavity, or cervix are all permissible).
- **3.2.6** Severe, active co-morbidity, defined as follows:
  - Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months prior to registration
  - Transmural myocardial infarction within the last 6 months prior to registration
  - History of stroke or transient ischemic attack within 6 months prior to registration.
  - Significant vascular disease (e.g., aortic aneurysm, history of aortic dissection) or clinically significant peripheral vascular disease.
  - Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
  - Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration
  - Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects; note, however, that laboratory tests for liver function other than screening panel (<u>Section 3.1</u>) and coagulation parameters are not required for entry into this protocol.
  - Acquired Immune Deficiency Syndrome (AIDS) based upon current CDC definition; note, however, that HIV testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive. Protocol-specific requirements may also exclude immuno-compromised patients.
- **3.2.7** Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the treatment involved in this study may be significantly teratogenic.
- **3.2.8** Prior allergic reaction to the study drug (Bevacizumab)
- **3.2.9** Prior history of hypertensive crisis or hypertensive encephalopathy.
- **3.2.10** History of a non-healing wound, ulcer, or bone fracture within 90 days (3 months) prior to registration
- **3.2.11** Gastrointestinal bleeding or any other hemorrhage/bleeding event CTCAE, v. 4 grade 3 or greater within 30 days prior to registration
- **3.2.12** Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to registration (with the exception of craniotomy)

## 4.0 PRETREATMENT EVALUATIONS/MANAGEMENT

NOTE: This section lists baseline evaluations needed <u>before the initiation of protocol treatment</u> that do not affect eligibility.

- **4.1** Highly Recommended Evaluations (4/15/14)
- **4.1.1** Baseline MR diffusion and perfusion imaging is optional but strongly recommended as further confirmation that the GTV is related to tumor and not radiation effect. The same type of enhanced

scan, i.e., MRI or CT, should be used throughout the period of protocol treatment for tumor measurement. See also Section 11.1.3.

- **4.1.2** The MGMT methylation status as a predictor of outcome will be obtained for the following patient groups:
  - Patients who have already had MGMT performed prior to registration into an /NRG Oncology/ RTOG GBM trial collecting MGMT methylation status.
  - Patients who have had MGMT analysis performed as routine care by a treating physician outside of an NRG Oncology/ RTOG GBM trial.
- **4.1.3** Pre-operative contrast-enhanced MRI or CT scan.

#### **5.0 REGISTRATION PROCEDURES** (10/9/14)

#### **Access requirements for OPEN and TRIAD:**

Site staff will need to be registered with CTEP and have a valid and active CTEP-IAM account. The Cancer Therapy Evaluation Program (CTEP) Identity and Access Management (IAM) application is a web-based application intended for use by both Investigators (i.e., all physicians involved in the conduct of NCI-sponsored clinical trials) and Associates (i.e., all staff involved in the conduct of NCI-sponsored clinical trials). Associates will use the CTEP-IAM application to register (both initial registration and annual re-registration) with CTEP and to obtain a user account.

Investigators will use the CTEP-IAM application to obtain a user account only. (See CTEP Investigator Registration Procedures below for information on registering with CTEP as an Investigator, which must be completed before a CTEP-IAM account can be requested.)

An active CTEP-IAM user account will be needed to access all CTEP and CTSU (Cancer Trials Support Unit) websites and applications, including the CTSU members' website.

Additional information can be found on the CTEP website at <a href="http://ctep.cancer.gov/branches/pmb/associate\_registration.htm">http://ctep.cancer.gov/branches/pmb/associate\_registration.htm</a>. For questions, please contact the *CTEP Associate Registration Help Desk* by email at <a href="mailto:ctepreghelp@ctep.nci.nih.gov">ctepreghelp@ctep.nci.nih.gov</a>.

<u>Note</u>: As of Amendment 1 activation, this trial is not utilizing the services of the ITC for dosimetry digital treatment data submission. See below for information on installing TRIAD for submission of digital RT data prior to enrolling patients.

## 5.1 Pre-Registration Requirements for Image-Guided Radiotherapy (IGRT) Treatment Approach (11/20/13)

**5.1.1** Institutions that plan to utilize PTV margins of less than 5 mm will also be required to complete image-guided radiotherapy (IGRT) credentialing for brain.

In order to utilize IGRT for margin reduction (see <u>Section 6.3</u>), the center must be credentialed for its use. This means the institution must have met technology requirements and have provided the baseline physics information. This information is available on the NRG Oncology/RTOG website, http://www.rtog.org/ClinicalTrials/ProtocolTable/StudyDetails.aspx?study=1205.

In order to become credentialed for brain IGRT, the institution must have already become credentialed for either 3DCRT and/or IMRT. Institutions that have not been credentialed by NRG Oncology to perform 3DCRT and/or IMRT MUST apply for 3DCRT and/or IMRT credentialing as described below in  $\underline{\text{Sections 5.2}}$  and  $\underline{\text{5.3}}$ .

## **5.1.2** *IGRT Credentialing Process*

- IGRT credentialing for brain (review of at least one case) will be required for institutions utilizing PTV margins of less than 5 mm (See Section 6.3). The first step is for the institution or investigator to update or complete a new Facility Questionnaire and/or set up an SFTP account for digital data submission. See Sectio 12 for details.
- Next, the institution must submit a series of daily treatment images along with a spreadsheet of IGRT data from an anonymized brain cancer patient. This information is available on the

on the NRG Oncology/RTOG website, <a href="http://www.rtog.org/ClinicalTrials/ProtocolTable/StudyDetails.aspx?study=1205">http://www.rtog.org/ClinicalTrials/ProtocolTable/StudyDetails.aspx?study=1205</a>. This series must include a minimum of 5 daily pre-treatment images obtained on sequential treatment days. Pre-treatment images may include three-dimensional (3D) volumetric images (either fan- or cone-beam CT with Megavoltage (MV) or kilovoltage (kV) x-ray or Orthogonal (MV or kV) 2D images. These images and the spreadsheet will be reviewed by the Study Chair, Christina Tsien, MD, and the Medical Physics Co-chair, Martha Matuszak, PhD, prior to certification.

## 5.2 Pre-Registration Requirements for IMRT Treatment Approach (2/27/14)

5.2.1 In order to utilize IMRT on this study (this includes all CyberKnife treatments), the institution must have met specific technology requirements and have provided baseline physics information. Instructions for completing these requirements or determining if they already have been met are available on the IROC Houston [formerly the Radiological Physics Center (RPC) web site]. Visit <a href="http://irochouston.mdanderson.org">http://irochouston.mdanderson.org</a> and select "Credentialing" and "Credentialing Status Inquiry".

An IMRT phantom study with the IROC Houston must be successfully completed (if the institution has not previously met this IMRT credentialing requirement). Instructions for requesting and irradiating the phantom are available on the IROC Houston web site at <a href="http://irochouston.mdanderson.org">http://irochouston.mdanderson.org</a>; select "Credentialing" and "RTOG". Upon review and successful completion of the phantom irradiation, IROC Houston will notify both the registering institution and NRG Oncology that the institution has completed this requirement. Subsequently, NRG Oncology will update the RSS database.

5.2.2 The institution or investigator must update or complete the electronic Facility Questionnaire (available on the IROC Houston web site at <a href="http://irochouston.mdanderson.org">http://irochouston.mdanderson.org</a>) and then complete a credentialing status inquiry form, also found on the IROC Houston, web site to determine if your site has met all of the requirements. This will be completed in place of updating the previous Facility Questionnaire. When the requirements are met, the site and NRG Oncology will be notified. NRG Oncology will then update the RSS database. Before any cases can be entered, a TRIAD account must also have been set up for data submission.

#### 5.3 Pre-Registration Requirements for 3D-CRT Treatment Approach (2/27/14)

- **5.3.1** Only institutions that have met the technology requirements and that have provided the baseline physics information that are described in 3D-CRT Quality Assurance Guidelines may enter patients onto this study.
- 5.3.2 The institution or investigator must update or complete a Facility Questionnaire (available on the RPC web site at http://irochouston.mdanderson.org) and complete a credentialing status inquiry form also found on the IROC Houston web site to determine if your site has met all of the requirements. This will be completed in place of updating the previous Facility Questionnaire. When the requirements are met the site and NRG Oncology will be notified. NRG Oncology will then update the RSS database prior to entering any cases. A TRIAD account must also have been set up for data submission prior to submitting any data. IROC Houston will notify the institution and NRG Oncology when all requirements have been met and the institution is eligible to enter patients onto this study. NRG Oncology will update the RSS database.

## 5.4 Pre-Registration Requirements for Proton Treatment Approach (2/27/14)

#### **5.4.1** Proton Credentialing Process

Proton therapy may be used on this protocol. Investigators using proton therapy must comply with the NCI proton guidelines for the Use of Proton Radiation Therapy in NCI Sponsored Cooperative Group Clinical Trials, which are available on the websites of the IROC Houston (<a href="http://irochouston.mdanderson.org">http://irochouston.mdanderson.org</a>), ATC (<a href="http://atc.wustl.edu">http://www.qarc.org</a>). These requirements include, but are not limited to, completion of a proton facility questionnaire, a successful IROC Houston site visit, which identifies the proton technique(s) which can be used, annual monitoring of the proton beam calibration, e.g. IROC Houston's monitoring program.

**5.4.2** Dose will be reported in Gy (RBE), where 1 Gy(RBE) = proton dose Gy x RBE (radiobiological effective dose), RBE = 1.1.

- **5.4.3** Radiation doses shall be prescribed using the protocol specified definitions for GTV and CTV. For set-up uncertainties and target motion, additional margin (including proximal and distal), smearing, and range of modulation will be added on a per beam basis. Proton treatment plans will be based upon a CT scanner for which the institution has defined an imaging protocol for protons which establishes the relationship between the CT number and the stopping power ratios.
- 5.4.4 The IROC Houston will coordinate the completion of the proton therapy use approval process in conjunction with the appropriate other Quality Assurance Offices for any additional protocol specific credentialing requirements. IROC Houston will notify the institution and NRG Oncology when all requirements have been met and the institution is eligible to enter patients onto this study. NRG Oncology will update the RSS database.
- **5.4.5** Additional credentialing requirements for this protocol may be found on the IROC Houston web site (http://irochouston.mdanderson.org) by selecting "Credentialing" and "RTOG".
- **5.4.6** Proton resources for this protocol include:

Michael T. Gillin, PhD Professor The University of Texas MD Anderson Cancer Center Department of Radiation Physics 713-563-2507/Fax: 713-563-2545 mgillin@mdanderson.org

Anita Mahajan, MD University of Texas MD Anderson Cancer Center 1515 Holcombe Boulevard Houston, TX 77030 713-563-2350 amahajan@mdanderson.org

5.4.7 If protons are to be used, review and successful completion of the "Dry-Run" QA test using protons is required, the IROC Houston will notify both the registering institution and NRG Oncology that the institution has successfully completed this requirement for protons

There are no proton protocol specific credentialing requirements for this protocol.

## 5.5 Digital RT Data Submission Using TRIAD (11/20/13)

TRIAD is the American College of Radiology's (ACR) image exchange application. TRIAD provides sites participating in RTOG clinical trials a secure method to transmit DICOM RT and other objects. TRIAD anonymizes and validates the images as they are transferred.

#### **TRIAD Access Requirements**

- Site physics staff who will submit images through TRIAD will need to be registered with The Cancer Therapy Evaluation Program (CTEP) and have a valid and active CTEP Identity and Access Management (IAM) account. Please refer to <u>Section 5.0</u> of the protocol for instructions on how to request a CTEP-IAM account.
- To submit images, the site physics user must have been assigned the 'TRIAD site user' role on the relevant Group or CTSU roster.
- RAs are able to submit standard of care imaging through the same method.

#### TRIAD Installations

When a user applies for a CTEP-IAM account with proper user role, he/she will need to have the TRIAD application installed on his/her workstation to be able to submit images. TRIAD installation documentation can be found on the NRG Oncology/RTOG website Core lab tab.

This process can be done in parallel to obtaining your CTEP IAM account username and password.

If you have any questions regarding this information, please send an email to the TRIAD Support mailbox at <a href="mailto:TRIAD-Support@acr.org">TRIAD-Support@acr.org</a>.

## 5.6 Regulatory Pre-Registration Requirements (10/9/14) Investigator Registration Requirements

Prior to the recruitment of a patient for this study, investigators must be registered members of a Lead Protocol Organization. Food and Drug Administration (FDA) regulations and National Cancer Institute (NCI) policy require all investigators participating in any NCI-sponsored clinical trial to register and to renew their registration annually. Registration requires the submission of:

- a completed **Statement of Investigator Form** (FDA Form 1572) with an original signature
- a current Curriculum Vitae (CV)
- a completed and signed Supplemental Investigator Data Form (IDF)
- a completed *Financial Disclosure Form* (FDF) with an original signature

Fillabe PDF forms and additional information can be found on the CTEP website at <a href="http://ctep.cancer.gov/investigatorResources/investigator\_registration.htm">http://ctep.cancer.gov/investigatorResources/investigator\_registration.htm</a>. For questions, please contact the *CTEP Investigator Registration Help Desk* by email at <a href="mailto:cpmbregpend@ctep.nci.nih.gov">cpmbregpend@ctep.nci.nih.gov</a>.

#### Site Registration Requirements [Insert as appropriate]

This study is supported by the NCI Cancer Trials Support Unit (CTSU).

### IRB Approval

Each investigator or group of investigators at a clinical site must obtain IRB approval for this protocol and submit IRB approval and supporting documentation to the CTSU Regulatory Office before they can be approved to enroll patients. Study centers can check the status of their registration packets by querying the Regulatory Support System (RSS) site registration status page of the CTSU members' website by entering credentials at <a href="https://www.ctsu.org">https://www.ctsu.org</a>.

#### **Downloading Site Registration Documents:**

Site registration forms may be downloaded from the *RTOG 1205* protocol page located on the CTSU members' website. Permission to view and download this protocol and its supporting documents is restricted and is based on person and site roster assignment housed in the CTSU RSS.

- Go to <a href="https://www.ctsu.org">https://www.ctsu.org</a> and log in to the members' area using your CTEP-IAM username and password
- Click on the Protocols tab in the upper left of your screen
- Click on the NRG Oncology link to expand, then select trial protocol #RTOG-1205.
- Click on the Site Registration Documents link

### Requirements RTOG 1205 Site Registration:

- CTSU IRB Certification CTSU IRB/Regulatory Approval Transmittal Sheet
- IRB Approval Letter
- IRB/REB Approved Informed Consent (English and native language versions\*) \*Note: Institutions must provide certification/verification of IRB/REB consent translation to NRG Headquarters (described below).
- IRB/REB registration number renewal information as appropriate.
- CTSU RT Facilities Inventory Form
   NOTE: Per NCI policy all institutions that participate on protocols with a radiation therapy component must participate in the Imaging and Radiation Oncology Core (IROC)

monitoring program. If this form has been previously submitted to CTSU it does not need to be resubmitted unless updates have occurred at the RT facility

## **Submitting Regulatory Documents:**

Submit completed forms along with a copy of your IRB Approval and Informed Consent to the CTSU Regulatory Office, where they will be entered and tracked in the CTSU RSS.

CTSU Regulatory Office

1818 Market Street, Suite 1100

Philadelphia, PA 19103 Phone: 1-866-651-2878 Fax: 215-569-0206

E-mail: CTSURegulatory@ctsu.coccq.org (for regulatory document submission only)

### **Checking Your Site's Registration Status:**

Check the status of your site's registration packets by querying the RSS site registration status page of the members' section of the CTSU website. (Note: Sites will not receive formal notification of regulatory approval from the CTSU Regulatory Office.)

- Go to <a href="https://www.ctsu.org">https://www.ctsu.org</a> and log in to the members' area using your CTEP-IAM username and password
- Click on the Regulatory tab at the top of your screen
- Click on the Site Registration tab
- Enter your 5-character CTEP Institution Code and click on Go

### Non-English Speaking Canadian and Non-North American Institutions

Translation of documents is critical. The institution is responsible for all translation costs. All regulatory documents, including the IRB/REB approved consent, must be provided in English and in the native language. Certification of the translation is optimal but due to the prohibitive costs involved NRG Oncology will accept, at a minimum, a verified translation. A verified translation consists of the actual REB approved consent document in English and in the native language, along with a cover letter on organizational/letterhead stationery that includes the professional title, credentials, and signature of the translator as well as signed documentation of the review and verification of the translation by a neutral third party. The professional title and credentials of the neutral third party translator must be specified as well.

#### **5.6.3** Pre-Registration Requirements FOR CANADIAN INSTITUTIONS

Prior to clinical trial commencement, Canadian institutions must complete and fax (215-569-0206) or e-mail (<a href="mailto:CTSURegulatory@ctsu.coccg.org">CTSURegulatory@ctsu.coccg.org</a>) the following Health Canada forms to the CTSU Regulatory Office:

- Health Canada's Therapeutic Products Directorates' Clinical Trial Site Information Form,
- Qualified Investigator Undertaking Form, and
- Research Ethics Board Attestation Form.

#### 5.6.4 Pre-Registration Requirements FOR INTERNATIONAL INSTITUTIONS

## • For institutions that do not have an approved LOI for this protocol:

International sites must submit an LOI to NRG Oncology to receive approval to participate in this trial. For more details see link below:

http://www.rtog.org/Researchers/InternationalMembers/LetterofIntent.aspx.

#### • For institutions that have an approved LOI for this protocol:

All requirements indicated in your LOI Approval Notification must be fulfilled prior to enrolling patients to this study.

#### **5.7 Registration** (10/9/14)

## **5.7.1** OPEN Registration Instructions

Patient registration can occur only after evaluation for eligibility is complete, eligibility criteria have been met, and the study site is listed as 'approved' in the CTSU RSS. Patients must have signed and dated all applicable consents and authorization forms.

Patient enrollment will be facilitated using the Oncology Patient Enrollment Network (OPEN). OPEN is a web-based registration system available on a 24/7 basis. To access OPEN, the site must have an active CTEP-IAM account (check at < https://eappsctep.nci.nih.gov/iam/index.jsp >) and a 'Registrar' role on either the LPO or participating organization roster. All site staff will use OPEN to enroll patients to this study. OPEN can be accessed at https://open.ctsu.org or from the OPEN tab on the CTSU members' web site https://www.ctsu.org.

Prior to accessing OPEN site staff should verify the following:

- All eligibility criteria have been met within the protocol stated timeframes. Site staff should
  use the registration forms provided on the group or CTSU web site as a tool to verify
  eligibility.
- All patients have signed an appropriate consent form and HIPAA authorization form (if applicable).

Further instructional information is provided on the OPEN tab of the CTSU members' side of the CTSU website at <a href="https://www.ctsu.org">https://www.ctsu.org</a> or at <a href="https://open.ctsu.org">https://open.ctsu.org</a>. For any additional questions contact the CTSU Help Desk at 1-888-823-5923 or <a href="ctsucontact@westat.com">ctsucontact@westat.com</a>.

5.7.2 In the event that the OPEN system is not accessible, participating sites can contact web support for assistance with web registration: <a href="websupport@acr.org">websupport@acr.org</a> or call the Registration Desk at (215) 574-3191, Monday through Friday, 8:30 a.m. to 5:00 p.m. ET. The registrar will ask the site to fax in the eligibility checklist and will need the registering individual's e-mail address and/or return fax number. This information is required to assure that mechanisms usually triggered by the OPEN web registration system (e.g. drug shipment and patient-specific calendar) will occur.

#### **6.0 RADIATION THERAPY** (11/20/13)

Note: Intensity Modulated RT (IMRT) Is Allowed.

Protons are permitted for institutions which have been approved and credentialed for protons, as protons may reduce the volume of normal tissue which will be re-irradiated. (If protons are used, to avoid delays resulting from unplanned equipment availability, photon therapy may be administered instead of proton therapy.)

<u>Note</u>: As of Amendment 1 activation, this trial is not utilizing the services of the ITC for dosimetry digital treatment data submission. See <u>Section 5</u> for information on installing TRIAD for submission of digital RT data PRIOR to enrolling patients.

#### 6.1 Dose Specifications

- **6.1.1** Photons: Treatment shall consist of 35 Gy delivered in 10 fractions. Target coverage and homogeneity limits and deviations are listed in Table 1.
- 6.1.2 Protons Absorbed dose: Doses are expressed in units of RBE-weighted absorbed dose, D<sub>RBE</sub>. For protons the RBE is taken to be 1.1. D<sub>RBE</sub> = 1.1 x D, where D represents the absorbed dose in Gy. Treatment shall consist of 35 Gy(RBE) delivered in 10 fractions. Target coverage and homogeneity limits and deviations are listed in Table 1.

Table 1. Target Coverage and Dose Limits

| Dose Metric | Per Protocol | Variation Acceptable | Deviation Unacceptable |
|---|---|---|---|
| Volume of PTV covered | Greater than or equal | Greater than or equal | Less than 90% of the |
| by the prescription dose | to 95% of the PTV | to 90% of the PTV | PTV receiving greater |
| photons 35 Gy – | should receive greater | receiving greater than | than or equal to photons |
| protons 35 Gy(RBE) | than or equal to | or equal to photons 35 | 35 Gy – protons 35 |
| | photons 35 Gy – | Gy – protons 35 | Gy(RBE) |
| | protons 35 Gy(RBE) | Gy(RBE) | |
| Minimum dose to the | Greater than or equal | Greater than or equal | Less than 28 Gy (80% of |
| PTV (0.03 cc) | to 29.75 Gy (85% of | to 28 Gy (80% of the | the prescription dose) – |

| | the prescription dose) – protons 29.75 Gy(RBE) | prescription dose) – protons 28 Gy(RBE); Minimum doses of less than 28 Gy are acceptable if they occur due to OAR/PTV overlap | protons 28 Gy(RBE);<br>Minimum doses of less<br>than 28 Gy are<br>unacceptable unless they<br>occur in regions of<br>OAR/PTV overlap |
|---|---|---|---|
| Maximum dose to the PTV (0.03 cc) | Less than or equal to<br>42 Gy (120% Rx<br>Dose) – protons 42<br>Gy(RBE) | Less than or equal to<br>45.50 Gy (130% Rx<br>Dose) – protons 45.50<br>Gy(RBE) | Greater than 45.50 Gy<br>(130% Rx Dose) –<br>protons 45.50 Gy(RBE) |

#### 6.2 Technical Factors [Equipment, energies]

The 10 treatment fractions of 3.5 Gy each will be delivered on consecutive treatment days (typically 5 fractions per week). Any FDA cleared external beam radiation delivery system may be used (including conventional linear accelerators, cyberknife systems, tomotherapy, proton therapy, etc.). Imaging for treatment planning will be obtained with the patient in the same position and immobilization device as for treatment. All patients will be positioned via a combination of rigid immobilization and daily image guidance to ensure positioning accuracy of 3 mm or better, and of a magnitude that justifies the PTV margin applied (the participating institutions must document the immobilization and localization methods applied).

#### 6.3 Localization, Simulation, and Immobilization (10/9/14)

An MRI and/or CT scanning obtained with the patient immobilized in the treatment position is , required for treatment planning. The image resolution of no worse than 1.5 mm x1.5 mm x 3 mm. Immobilization must be rigid (e.g. thermoplastic masks). For daily treatment, localization will include the steps of a) immobilization with the same device used for simulation, and b) daily image guidance using at a minimum orthogonal pairs of radiographs aligned to DRRs as a computer-assisted process (CT-CBCT alignment is permitted as well). Institutions utilizing PTV margins of less than 5 mm are required to undergo IGRT credentialing for brain (see Section 5.1).

## **6.4** Treatment Planning/Target Volumes (10/9/14)

A GTV will be defined using contrast-enhanced CT and/or MRI images. The post-operative resection cavity will be outlined if no residual enhancing tumor is noted. A CTV expansion of no more than 5 mm is optional for lesions measuring less than 3.5 cm in maximum diameter or if this is a new lesion, but must be reported when used. Otherwise, no additional CTV expansion will be added. A PTV expansion that is justified based on image guidance and immobilization will be applied. Regardless of immobilization and localization methods, the PTV expansion should be no smaller than 3 mm. As noted in Section 6.3, institutions utilizing PTV margins of less than 5 mm are required to undergo IGRT credentialing for brain (see Section 5.1) and utilize computer-assisted daily IGRT for all treatment fractions.

If protons are used, an adjustment must be made within the treatment planning process to take into account of range uncertainties along the beam direction, following the established practice at the specific proton facility, which should be based on the recommendations contained in ICRU 78, paragraph 5.1.4.4.

Treatment planning using multiple, non-coplanar beams or arc-based therapy is advised. IMRT based planning is allowed. To ensure dose calculation accuracy, the minimum field size used should be consistent with the minimum field size commissioned for use at the institution and should not be smaller than 2 cm x 2 cm. In any case, the objective of treatment planning is to ensure sufficient dose conformity that the normal tissue constraints are met.

### 6.5 Critical Structures (2/27/14)

Normal tissues to be contoured will include the brain, brainstem, optic nerves and chiasm. Planning risk volume (PRV) expansions (minimum of 3 mm) should be utilized for optic nerves

and chiasm. Special consideration should be given to avoid doses greater than the prescription dose within the scalp as well as limiting the exit dose through the oral cavity and mucosa. The treatment parameters should be modified to optimize the conformity of the prescription isodose volume to the target volume while minimizing dose to critical structures. There are two scenarios for normal tissues limits: (1) previous radiation to the local area including critical organs at risk and (2) no previous radiation to the local area or organs at risk. The limits for both scenarios are given in Table 2.

Table 2. Normal Tissue Dose Limits

| Dose Metric | Per Protocol | Variation Acceptable | Deviation Unacceptable |
|---|---|---|---|
| Scenario (1): Previous radiation | Scenario (1): Previous radiation to the local area including critical organs at risk | | |
| Maximum Dose to PRV for Optic Nerves and Chiasm (0.03 cc) | Less than or equal to<br>20 Gy photons – 20<br>Gy(RBE) protons | Greater than 20 Gy<br>but less than or equal<br>to 25 Gy photons –<br>25 Gy(RBE) protons | Greater than 25 Gy<br>photons – 25 Gy(RBE)<br>protons |
| Maximum Dose to Brainstem (0.03 cc) | Less than or equal to<br>24 Gy photons – 24<br>Gy(RBE) protons | Greater than 24 Gy<br>but less than or equal<br>to 30 Gy photons –<br>30 Gy(RBE) protons | Greater than 30 Gy<br>photons – 30 Gy(RBE)<br>protons |
| Scenario (2): No previous radia | tion to the local area o | r critical organs at risk | |
| Maximum Dose to PRV for<br>Optic Nerves and Chiasm (0.03<br>cc) | Less than or equal to<br>35 Gy (the<br>prescription dose)<br>photons – 35<br>Gy(RBE) protons | Greater than 35 Gy<br>but less than or equal<br>to 36.75 Gy (105 % of<br>the prescription dose)<br>photons – 36.75<br>Gy(RBE) protons | Greater than 36.75 Gy<br>(105% of the prescription<br>dose) photons – 36.75<br>Gy(RBE) protons |
| Maximum Dose to Brainstem (0.03 cc) | Less than or equal to<br>35 Gy (the<br>prescription dose)<br>photons – 35<br>Gy(RBE) protons | Greater than 35 Gy<br>but less than or equal<br>to 36.75 Gy (105 % of<br>the prescription dose)<br>photons – 36.75<br>Gy(RBE) protons | Greater than 36.75 Gy<br>(105 % of the<br>prescription dose)<br>photons – 36.75<br>Gy(RBE) protons |

#### 6.5.1 Standard Structure Names for TRIAD Submission

All structures must be submitted and labeled according to the specifications in the table below or resubmission will be required.

| Standard Name | Description | Reference Dose (GY) | Validation Profile |
|---|---|---|---|
| GTV_3500 | Residual enhancing tumor or post-operative resection cavity | 35 | Required |
| CTV_3500 | An Optional CTV expansion of no more than 5 mm. | 35 | Required |
| PTV_3500 | planning target volume; an additional margin of 3 to 5 mm | 35 | Required |
| Brain | Outline of the brain | | Required |
| OpticChiasm | Optic Chiasm | | Required |
| OptChiasm_PRV | Optic Chiasm Planning Risk Volume | | Required |
| BrainStem | Brain Stem | | Required |
| BrainStem_PRV | Brain Stem Planning Risk Volume | | Required |

| OpticNerve_L | Left Optic Nerve | Required |
|--------------|-------------------------------------------|----------|
| OptNrv_L_PRV | Left Optic Nerve Planning<br>Risk Volume | Required |
| OpticNerve_R | Right Optic Nerve | Required |
| OptNrv_R_PRV | Right Optic Nerve Planning<br>Risk Volume | Required |

#### 6.6 Documentation Requirements

At the completion of treatment, the following should be forwarded to NRG Oncology: daily treatment record and the radiotherapy summary per <u>Section 12.1</u>. In addition, CT/MRI documentation must be submitted per <u>Section 12.2</u>. Isodose distributions should be displayed on orthogonal planes or, if not possible, on multiple transverse slices through each target.

#### 6.7 Compliance Criteria

See Tables 1 and 2 for target and normal tissue compliance criteria.

#### 6.8 R.T. Quality Assurance Reviews

The Radiation Oncology Co-Chair, Christina Tsien, M.D., will perform an RT Quality Assurance Review of cases on an ongoing basis. The final cases will be reviewed within 6 months after this study has reached the target accrual or as soon as complete data for all cases enrolled has been received at Imaging and Radiation Oncology Core (IROC) Philadelphia, whichever occurs first. These reviews will be ongoing and performed at the NRG Oncology semi-annual meetings as well as at IROC Philadelphia.

#### 6.9 Radiation Therapy Adverse Events

#### **6.9.1** Acute

Expected acute radiation-induced toxicities include hair loss, fatigue, and erythema or soreness of the scalp. Potential acute toxicities include nausea and vomiting as well as temporary aggravation of brain tumor symptoms such as headaches, seizures, and weakness. Reactions in the ear canals and on the ear should be observed and treated symptomatically; these reactions could result in short-term hearing impairment. Dry mouth or altered taste have been occasionally reported.

#### 6.9.2 Early Delayed

Possible early delayed radiation effects include lethargy and transient worsening of existing neurological deficits occurring 1-3 months after radiotherapy treatment.

#### **6.9.3** Late Delayed

Possible late delayed effects of radiotherapy include risk of radiation necrosis, and endocrine dysfunction. In addition, neurocognitive deficits, which could lead to mental slowing and behavioral change, are possible. Permanent hearing impairment and visual damage are rare. Cataracts can be encountered.

### 6.10 Radiation Therapy Adverse Event Reporting

See Section 7.6.

#### 7.0 DRUG THERAPY

Protocol treatment must begin within 14 days after registration.

#### **7.1** Treatment (10/9/14)

#### **7.1.1** Dose Definition

.Bevacizumab will be administered at a dose of 10 mg/kg every 2 weeks. The patient's weight must be checked prior to each dose of bevacizumab. Doses will be adjusted if there is a > 10% change in weight.

#### **7.1.2** Technique of Administration

Bevacizumab will be administered intravenously per institutional guidelines with associated premedications.

## 7.1.3 <u>Duration of Treatment</u>

Initial cycle of bevacizumab must start within 14 days of registration. A deviation of  $\pm$ -3 days is permitted. If beyond this timing period, the imaging and work-up will need to be repeated. Subsequent bevacizumab doses may be given every 14 days apart  $\pm$ -3 days due to holidays, etc. Treatment may be held for  $\pm$  grade 3 toxicities as defined in Section 7.3.

**Arm 1**: Patients randomized to the bevacizumab alone arm will be administered bevacizumab every 2 weeks until disease progression.

**Arm 2**: Patients randomized to the bevacizumab and re-irradiation arm will receive an initial induction dose of bevacizumab (alone without radiation). It will then be followed by concurrent bevacizumab and radiation at the next dose which is administered 14 days later. This will allow additional time for radiation therapy planning especially in symptomatic patients. Concurrent bevacizumab cycle may be given either on the day prior to start of radiation or on day 1 of radiation. Bevacizumab will then be continued every 2 weeks until disease progression.

#### **7.2** Bevacizumab Agent Information (10/3/16)

Consult the package insert for detailed pharmacologic and safety information.

## 7.2.1 Description and Packaging

Bevacizumab is a humanized IgG1 monoclonal antibody (MAb) that binds all biologically active isoforms of human VEGF (or VEGF-A) with high affinity (kd = 1.1 nM). The antibody consists of a human IgG1 framework and the antigen-binding complementarity-determining regions from the murine anti-VEGF MAb A.4.6.1.16-18. Vials contain bevacizumab with phosphate, trehalose, polysorbate 20, and sterile water for injection (SWFI), USP.

#### **7.2.2** Administration

Bevacizumab should be administered as a continuous intravenous infusion using a rate-regulating device per institutional guidelines with associated pre-medications. Do not administer as an IV push or bolus. If no institutional guidelines exist, follow below:

Administer the initial dose over a minimum of 90 minutes. If no adverse reactions occur, administer the second dose over a minimum of 60 minutes. If no adverse reactions occur after the second dose, administer subsequent doses over a minimum of 30 minutes. If infusion-related adverse reactions occur, all subsequent infusions should be administered over the shortest period that was well tolerated.

#### **7.2.3** Storage

Vials contain no preservative and are suitable for single use only.

### **7.2.4** Supply

Commercially available.

#### Non-Canadian International Institutions

Please refer to your LOI Approval Notification. Your institution will be responsible for acquiring any drug noted in the protocol as commercially available and not provided for the study.

#### **7.2.5** Adverse Events

# Comprehensive Adverse Events and Potential Risks list (CAEPR) for Bevacizumab (rhuMAb VEGF, NSC 704865)

The Comprehensive Adverse Event and Potential Risks list (CAEPR) provides a single list of reported and/or potential adverse events (AE) associated with an agent using a uniform presentation of events by body system. In addition to the comprehensive list, a subset, the Specific Protocol Exceptions to Expedited Reporting (SPEER), appears in a separate column and is identified with bold and italicized text. This subset of AEs (SPEER) is a list of events that are protocol specific exceptions to expedited reporting to NCI (except as noted below). Refer to the 'CTEP, NCI Guidelines: Adverse Event Reporting

Requirements' <a href="http://ctep.cancer.gov/protocolDevelopment/electronic\_applications/docs/aeguidelines.pdf">http://ctep.cancer.gov/protocolDevelopment/electronic\_applications/docs/aeguidelines.pdf</a> for further clarification. *Frequency is provided based on 3540 patients*. Below is the CAEPR for bevacizumab (rhuMAb VEGF).

**NOTE**: Report AEs on the SPEER <u>ONLY IF</u> they exceed the grade noted in parentheses next to the AE in the SPEER. If this CAEPR is part of a combination protocol using multiple investigational agents and has an AE listed on different SPEERs, use the lower of the grades to determine if expedited reporting is required.

Version 2.4, May 23, 2016<sup>1</sup>

| Adverse Events with Possible<br>Relationship to Bevacizumab (rhuMAb VEGF)<br>(CTCAE 4.0 Term)<br>[n= 3540] | | | Specific Protocol Exceptions to Expedited Reporting (SPEER) |
|---|---|---|---|
| Likely (>20%) | Less Likely (<=20%) | Rare but Serious (<3%) | |
| <b>BLOOD AND LYMPHATIC</b> | SYSTEM DISORDERS | | |
| | Anemia | | Anemia (Gr 3) |
| | Cobrillo no utropo o si o | Blood and lymphatic system disorders - Other (renal thrombotic microangiopathy) | Fabrila nautus nania (Or 2) |
| CARRIAC DICORDERC | Febrile neutropenia | | Febrile neutropenia (Gr 3) |
| CARDIAC DISORDERS | | | |
| | Cardiac disorders - Other (supraventricular arrhythmias) <sup>3</sup> | Acute coronary syndrome <sup>2</sup> | Cardiac disorders - Other<br>(supraventricular arrhythmias) <sup>3</sup> (Gr 3) |
| | | Heart failure | |
| | | Left ventricular systolic dysfunction | |
| | | Myocardial infarction <sup>2</sup> | |
| | | Ventricular arrhythmia | |
| | | Ventricular fibrillation | |
| GASTROINTESTINAL DIS | ORDERS | | |
| | Abdominal pain | | Abdominal pain (Gr 3) |
| | Colitis | | Colitis (Gr 3) |
| | Constipation | | Constipation (Gr 3) |
| | Diarrhea | | Diarrhea (Gr 3) |
| | Dyspepsia | | Dyspepsia (Gr 2) |
| | | Gastrointestinal fistula⁴ | |
| | Gastrointestinal hemorrhage <sup>5</sup> Gastrointestinal obstruction <sup>6</sup> | | Gastrointestinal hemorrhage⁵ (Gr 2) |
| | | Gastrointestinal perforation <sup>7</sup> Gastrointestinal ulcer <sup>8</sup> | |
| | lleus | Caca officoafficial dioci | |
| | Mucositis oral | | Mucositis oral (Gr 3) |
| | Nausea | | Nausea (Gr 3) |
| | Vomiting | | Vomiting (Gr 3) |
| GENERAL DISORDERS A | ND ADMINISTRATION SITI | = CONDITIONS | |
| | Fatigue | | Fatigue (Gr 3) |
| | Infusion related reaction | | Infusion related reaction (Gr 2) |
| | Non-cardiac chest pain | | Non-cardiac chest pain (Gr 3) |
| | Pain | | Pain (Gr 3) |
| HEPATOBILIARY DISORD | | | (51.5) |
| | | Gallbladder perforation | |

| Adverse Events with Possible Relationship to Bevacizumab (rhuMAb VEGF) (CTCAE 4.0 Term) [n= 3540] | | Specific Protocol Exceptions to Expedited Reporting (SPEER) | |
|---|---|---|---|
| Likely (>20%) | Less Likely (<=20%) | Rare but Serious (<3%) | |
| IMMUNE SYSTEM DISOR | DERS | | |
| | Allergic reaction | | Allergic reaction (Gr 2) |
| | | Anaphylaxis | |
| INFECTIONS AND INFEST | | | |
| | Infection <sup>9</sup> | | Infection <sup>9</sup> (Gr 3) |
| | | Infections and infestations - Other (necrotizing fasciitis) | |
| | Infections and infestations - Other (peri-rectal abscess) | | |
| INJURY, POISONING AND | PROCEDURAL COMPLIC | CATIONS | |
| | | Injury, poisoning and procedural complications - Other (anastomotic leak) <sup>10</sup> | |
| | Wound complication | | Wound complication (Gr 2) |
| | Wound dehiscence | | Wound dehiscence (Gr 2) |
| INVESTIGATIONS | | | |
| | Alanine aminotransferase increased | | Alanine aminotransferase increased (Gr 3) |
| | Alkaline phosphatase increased | | Alkaline phosphatase increased (Gr<br>3) |
| | Aspartate aminotransferase increased | | Aspartate aminotransferase increased (Gr 3) |
| | Blood bilirubin increased | | Blood bilirubin increased (Gr 2) |
| | Creatinine increased | | |
| Neutrophil count decreased | | | Neutrophil count decreased (Gr 3) |
| | Platelet count decreased | | Platelet count decreased (Gr 4) |
| | Weight loss | | Weight loss (Gr 3) |
| | White blood cell decreased | | White blood cell decreased (Gr 3) |
| METABOLISM AND NUTF | RITION DISORDERS | | |
| | Anorexia | | Anorexia (Gr 3) |
| | Dehydration | | Dehydration (Gr 3) |
| | Hyperglycemia | | |
| | Hypokalemia | | |
| | Hyponatremia | | |
| MUSCULOSKELETAL AN | D CONNECTIVE TISSUE D | DISORDERS | |
| | Arthralgia | | Arthralgia (Gr 3) |
| | | Avascular necrosis <sup>11</sup> | |
| | Generalized muscle weakness | | |
| | Musculoskeletal and connective tissue disorder - Other (bone metaphyseal dysplasia) <sup>12</sup> | | |
| | Myalgia | | Myalgia (Gr 3) |
| | Osteonecrosis of jaw <sup>13</sup> | 1 | |
| NERVOUS SYSTEM DISC | | <u></u> | |
| | Dizziness | 1 | Dizziness (Gr 2) |
| | Headache | | Headache (Gr 3) |
| | | Intracranial hemorrhage | |

| Adverse Events with Possible Relationship to Bevacizumab (rhuMAb VEGF) (CTCAE 4.0 Term) [n= 3540] | | Specific Protocol Exceptions to Expedited Reporting (SPEER) | |
|---|---|---|---|
| Likely (>20%) | Less Likely (<=20%) | Rare but Serious (<3%) | |
| | | Ischemia cerebrovascular <sup>2</sup> | |
| | Peripheral sensory neuropathy <sup>14</sup> | | |
| | | Reversible posterior leukoencephalopathy syndrome | |
| DENIAL AND LIDINA DV DI | Syncope | | |
| RENAL AND URINARY DI | SURDERS | 1 | |
| | I I a manata min | Acute kidney injury | Hamaturia (Cr. 2) |
| | Hematuria Proteinuria | | Hematuria (Gr 3)<br>Proteinuria (Gr 2) |
| | FIOLEIIIUIIA | Renal and urinary disorders | rioteiliulia (Gi 2) |
| | | - Other (nephrotic syndrome) | |
| | | Urinary fistula | |
| REPRODUCTIVE SYSTEM | M AND BREAST DISORDE | | |
| Reproductive system and breast disorders - Other (ovarian failure) <sup>15</sup> | | | |
| | | Vaginal fistula | |
| | Vaginal hemorrhage | | Vaginal hemorrhage (Gr 3) |
| RESPIRATORY, THORAC | CIC AND MEDIASTINAL DIS | SORDERS | |
| | Allergic rhinitis | | Allergic rhinitis (Gr 3) |
| | | Bronchopleural fistula | |
| | | Bronchopulmonary hemorrhage | |
| | Cough | | Cough (Gr 3) |
| | Dyspnea | | Dyspnea (Gr 2) |
| | Epistaxis | | Epistaxis (Gr 3) |
| | Hoarseness | Respiratory, thoracic and mediastinal disorders - Other (nasal-septal perforation) Respiratory, thoracic and mediastinal disorders - Other | |
| | | (tracheo-esophageal fistula) | |
| SKIN AND SUBCUTANEC | <del>\</del> | | |
| | Dry skin | | |
| | Erythroderma | Palmar-plantar<br>erythrodysesthesia<br>syndrome | |
| | Pruritus | | Pruritus (Gr 2) |
| | Rash maculo-papular | | Rash maculo-papular (Gr 2) |
| \(\(\alpha\) | Urticaria | | Urticaria (Gr 2) |
| VASCULAR DISORDERS | | | |
| Hypertension | Thromboembolic event | | Hypertension (Gr 3) Thromboembolic event (Gr 3) |

| Adverse Events with Possible Relationship to Bevacizumab (rhuMAb VEGF) (CTCAE 4.0 Term) [n= 3540] | | | Specific Protocol Exceptions to Expedited Reporting (SPEER) |
|---|---|---|---|
| Likely (>20%) | Less Likely (<=20%) | Rare but Serious (<3%) | |
| | | Vascular disorders - Other (arterial thromboembolic event) <sup>2,16</sup> | |

<sup>&</sup>lt;sup>1</sup>This table will be updated as the toxicity profile of the agent is revised. Updates will be distributed to all Principal Investigators at the time of revision. The current version can be obtained by contacting <a href="PIO@CTEP.NCI.NIH.GOV">PIO@CTEP.NCI.NIH.GOV</a>. Your name, the name of the investigator, the protocol and the agent should be included in the e-mail.

<sup>&</sup>lt;sup>2</sup>The risks of arterial thrombosis such as cardiac or CNS ischemia are increased in elderly patients and in patients with a history of diabetes.

<sup>&</sup>lt;sup>3</sup>Supraventricular arrhythmias may include supraventricular tachycardia, atrial fibrillation, and atrial flutter.

<sup>&</sup>lt;sup>4</sup>Gastrointestinal fistula may include: Anal fistula, Colonic fistula, Duodenal fistula, Esophageal fistula, Gastric fistula, Gastrointestinal fistula, Rectal fistula, and other sites under the GASTROINTESTINAL DISORDERS SOC.

<sup>&</sup>lt;sup>5</sup>Gastrointestinal hemorrhage may include: Colonic hemorrhage, Duodenal hemorrhage, Esophageal hemorrhage, Esophageal varices hemorrhage, Gastric hemorrhage, Hemorrhoidal hemorrhage, Intraabdominal hemorrhage, Oral hemorrhage, Rectal hemorrhage, and other sites under the GASTROINTESTINAL DISORDERS SOC.

<sup>&</sup>lt;sup>6</sup>Gastrointestinal obstruction may include: Colonic obstruction, Duodenal obstruction, Esophageal obstruction, Ileal obstruction, Jejunal obstruction, Rectal obstruction, Small intestinal obstruction, and other sites under the GASTROINTESTINAL DISORDERS SOC.

<sup>&</sup>lt;sup>7</sup>Gastrointestinal perforation may include: Colonic perforation, Duodenal perforation, Esophageal perforation, Gastric perforation, Jejunal perforation, Rectal perforation, and Small intestinal perforation.

<sup>&</sup>lt;sup>8</sup>Gastrointestinal ulcer may include: Duodenal ulcer, Esophageal ulcer, Gastric ulcer, and other sites under the GASTROINTESTINAL DISORDERS SOC.

<sup>&</sup>lt;sup>9</sup>Infection may include any of the 75 infection sites under the INFECTIONS AND INFESTATIONS SOC.

<sup>&</sup>lt;sup>10</sup>Anastomotic leak may include Gastric anastomotic leak; Gastrointestinal anastomotic leak; Large intestinal anastomotic leak; Rectal anastomotic leak; Small intestinal anastomotic leak; Urostomy leak; Vaginal anastomotic leak.

<sup>&</sup>lt;sup>11</sup>There have been reports of non-mandibular osteonecrosis (avascular necrosis) in patients under the age of 18 treated with bevacizumab.

<sup>&</sup>lt;sup>12</sup>Metaphyseal dysplasia was observed in young patients who still have active epiphyseal growth plates.

<sup>&</sup>lt;sup>13</sup>Cases of osteonecrosis of the jaw (ONJ) have been reported in cancer patients in association with bevacizumab treatment, the majority of whom had received prior or concomitant treatment with i.v. bisphosphonates.

<sup>&</sup>lt;sup>14</sup>Increased rate of peripheral sensory neuropathy has been observed in trials combining bevacizumab and chemotherapy compared to chemotherapy alone.

Adverse events reported on bevacizumab (rhuMAb VEGF) trials, but for which there is insufficient evidence to suggest that there was a reasonable possibility that bevacizumab (rhuMAb VEGF) caused the adverse event:

**BLOOD AND LYMPHATIC SYSTEM DISORDERS** - Blood and lymphatic system disorders - Other (idiopathic thrombocytopenia purpura); Bone marrow hypocellular; Disseminated intravascular coagulation; Hemolysis

**CARDIAC DISORDERS** - Atrioventricular block complete; Atrioventricular block first degree; Cardiac arrest; Myocarditis; Pericardial effusion; Restrictive cardiomyopathy; Right ventricular dysfunction **EAR AND LABYRINTH DISORDERS** - Ear and labyrinth disorders - Other (tympanic membrane perforation); Hearing impaired; Tinnitus; Vertigo

**ENDOCRINE DISORDERS** - Hyperthyroidism; Hypothyroidism

**EYE DISORDERS** - Blurred vision; Cataract; Dry eye; Extraocular muscle paresis; Eye disorders - Other (blindness); Eye disorders - Other (conjunctival hemorrhage); Eye disorders - Other (corneal epithelial defect); Eye disorders - Other (floaters); Eye disorders - Other (ischemic CRVO); Eye disorders - Other (macular pucker); Eye disorders - Other (transient increased IOP > or =30 mm Hg); Eye disorders - Other (vitreous hemorrhage); Eye pain; Keratitis; Optic nerve disorder; Photophobia; Retinal detachment; Retinal tear; Retinopathy; Watering eyes

**GASTROINTESTINAL DISORDERS** - Ascites; Chelitis; Colonic stenosis; Dry mouth; Dysphagia; Enterocolitis; Esophageal pain; Esophageal stenosis; Flatulence; Gastrointestinal disorders - Other (peritonitis); Oral pain; Pancreatitis; Proctitis; Rectal mucositis; Rectal stenosis; Typhlitis

**GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS** - Death NOS; Edema face; Edema limbs; Edema trunk; Facial pain; Fever; Flu like symptoms; Gait disturbance; Injection site reaction; Localized edema; Multi-organ failure; Sudden death NOS

**HEPATOBILIARY DISORDERS** - Cholecystitis; Gallbladder necrosis; Gallbladder obstruction; Hepatic failure; Hepatic necrosis

**INJURY, POISONING AND PROCEDURAL COMPLICATIONS** - Arterial injury; Bruising; Burn; Dermatitis radiation: Fracture

**INVESTIGATIONS** - Activated partial thromboplastin time prolonged; Blood antidiuretic hormone abnormal; CD4 lymphocytes decreased; CPK increased; Carbon monoxide diffusing capacity decreased; Electrocardiogram QT corrected interval prolonged; Forced expiratory volume decreased; GGT increased; INR increased; Lipase increased; Lymphocyte count decreased; Serum amylase increased; Weight gain

**METABOLISM AND NUTRITION DISORDERS** - Acidosis; Hypercalcemia; Hyperkalemia; Hypermagnesemia; Hypernatremia; Hypertriglyceridemia; Hyperuricemia; Hypoalbuminemia; Hypocalcemia; Hypomagnesemia; Hypophosphatemia

MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS - Arthritis; Back pain; Bone pain; Chest wall pain; Fibrosis deep connective tissue; Head soft tissue necrosis; Joint effusion; Muscle weakness lower limb; Musculoskeletal and connective tissue disorder - Other (aseptic necrotic bone); Musculoskeletal and connective tissue disorder - Other (myasthenia gravis); Musculoskeletal and connective tissue disorder - Other (polymyalgia rheumatica); Neck pain; Pain in extremity; Pelvic soft tissue necrosis; Soft tissue necrosis lower limb

**NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (INCL CYSTS AND POLYPS)** - Tumor pain **NERVOUS SYSTEM DISORDERS** - Arachnoiditis; Ataxia; Central nervous system necrosis; Cerebrospinal fluid leakage; Cognitive disturbance; Depressed level of consciousness; Dysesthesia;

<sup>&</sup>lt;sup>15</sup>Ovarian failure, defined as amenorrhea lasting 3 or more months with follicle-stimulating hormone (FSH) elevation (≥30 mIU/mL), was increased in patients receiving adjuvant bevacizumab plus mFOLFOX compared to mFOLFOX alone (34% vs. 2%). After discontinuation of bevacizumab, resumption of menses and an FSH level <30 mIU/mL was demonstrated in 22% (7/32) of these women. Long term effects of bevacizumab exposure on fertility are unknown.

<sup>&</sup>lt;sup>16</sup>Arterial thromboembolic event includes visceral arterial ischemia, peripheral arterial ischemia, heart attack, and stroke.

Dysgeusia; Dysphasia; Encephalopathy; Extrapyramidal disorder; Facial nerve disorder; Hydrocephalus; Leukoencephalopathy; Memory impairment; Nervous system disorders - Other (increased intracranial pressure); Paresthesia; Peripheral motor neuropathy; Pyramidal tract syndrome; Seizure; Somnolence; Tremor; Vasovagal reaction

**PSYCHIATRIC DISORDERS** - Agitation; Anxiety; Confusion; Depression; Insomnia; Libido decreased; Psychosis

**RENAL AND URINARY DISORDERS** - Bladder spasm; Chronic kidney disease; Cystitis noninfective; Renal and urinary disorders - Other (dysuria); Renal and urinary disorders - Other (ureterolithiasis); Renal hemorrhage; Urinary frequency; Urinary incontinence; Urinary retention; Urinary tract obstruction; Urinary tract pain

**REPRODUCTIVE SYSTEM AND BREAST DISORDERS** - Breast pain; Erectile dysfunction; Irregular menstruation; Pelvic pain; Vaginal discharge

**RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS** - Adult respiratory distress syndrome; Atelectasis; Hypoxia; Nasal congestion; Pulmonary fibrosis; Pulmonary hypertension; Respiratory failure; Respiratory, thoracic and mediastinal disorders - Other (dry nares); Respiratory, thoracic and mediastinal disorders - Other (pulmonary infarction)

**SKIN AND SUBCUTANEOUS TISSUÉ DISORDERS** - Alopecia; Hyperhidrosis; Nail loss; Pain of skin; Photosensitivity; Purpura; Rash acneiform; Skin and subcutaneous tissue disorders - Other (diabetic foot ulcer); Skin and subcutaneous tissue disorders - Other (skin breakdown/ decubitus ulcer); Skin hyperpigmentation; Skin induration; Skin ulceration; Stevens-Johnson syndrome

VASCULAR DISORDERS - Flushing; Hot flashes; Hypotension; Lymphocele; Phlebitis; Vasculitis

**Note**: Bevacizumab (rhuMAb VEGF) in combination with other agents could cause an exacerbation of any adverse event currently known to be caused by the other agent, or the combination may result in events never previously associated with either agent.

### **7.3 Bevacizumab Dose Modifications** (8/24/15)

**7.3.1** First dose: The dose of bevacizumab will be 10 mg/kg delivered intravenously. There will be no dose reduction for bevacizumab. Treatment should be interrupted or discontinued for certain adverse events, as described below. If bevacizumab is interrupted for ANY reason for > 8 weeks, the patient should discontinue bevacizumab therapy on protocol.

**Treatment Modification for Bevacizumab-Related Adverse Events** 

| Event | CTCAE.v4.0 Grade | Action To Be Taken |
|---|---|---|
| Allergic reactions | Grade 1-3 | If infusion-related or allergic reactions occur, premedications should be given with the next dose and infusion time may not be reduced for the subsequent infusion. Follow the |
| | | guidelines in Section 7.3 for bevacizumab administration. |
| Acute infusional reactions/<br>cytokine release syndrome | | For patients with grade 3 reactions, bevacizumab |
| Cytokine release Syndrome | | infusion should be stopped and not restarted on the same day. At the physicians' discretion, bevacizumab may be permanently discontinued or re-instituted with premedications and administered no faster than 60 minutes. If bevacizumab is re-instituted, the patient should be closely monitored for a duration comparable to or longer than the duration of the previous reactions. |
| | Grade 4 | Discontinue bevacizumab |
| Arterial Thrombosis | Grade 2 ( if new or<br>worsened since<br>bevacizumab therapy) | Discontinue bevacizumab |

| Event | CTCAE.v4.0 Grade | Action To Be Taken |
|---|---|---|
| CVA) - any peripheral or visceral arterial ischemia/thrombosis | Grade 3-4 | Discontinue bevacizumab |
| Venous Thrombosis | | |
| | Grade 3<br>OR<br>asymptomatic grade 4 | <ul> <li>Hold bevacizumab treatment. If the planned duration of full-dose anticoagulation is &lt; 2 weeks, bevacizumab should be held until the full-dose anticoagulation period is over.</li> <li>If the planned duration of full-dose anticoagulation is &gt;2</li> </ul> |
| | | weeks, bevacizumab may be resumed during the period of full-dose anticoagulation <b>IF</b> <u>all</u> of the criteria below are met: |
| | | <ul> <li>The subject must have an in-range INR (usually 2-3) on a stable dose of warfarin or be on a stable dose of heparin prior to restarting bevacizumab</li> <li>The subject must not have pathological conditions that carry high risk of bleeding (eg, tumor involving major vessels or other conditions)</li> <li>The subject must not have had hemorrhagic events while on study</li> </ul> |
| | | <ul> <li>If thromboemboli worsen/recur upon resumption of study<br/>therapy, discontinue bevacizumab</li> </ul> |
| | Grade 4 (symptomatic) | Discontinue bevacizumab |
| Hypertension* | [Treat with antihypertens consistent with general r | sive medication as needed. The goal of BP control should be medical practice] |
| | Grade 1 | Consider increased BP monitoring |
| | Grade 2 asymptomatic | Begin anti-hypertensive therapy and continue bevacizumab |
| | -Grade 2 symptomatic or Grade 3 | Hold bevacizumab until symptoms resolve AND BP < 160/100mmHg |
| | Grade 4 | Discontinue bevacizumab |
| Congestive Heart Failure | Grade 3 | Discontinue bevacizumab |
| | Grade 4 | Discontinue bevacizumab |
| Proteinuria | ratio before every dose of performed ] | nonitored by urine dipstick or urine protein creatinine (UPC) of bevacizumab, if dip is > 2 + then a UPC ratio should be |
| | UPC ratio<br>< 3.5 | Continue bevacizumab |
| | UPC ratio<br>≥ 3.5 | Hold bevacizumab until UPC recovers to < 3.5 |
| | Grade 4 or nephrotic syndrome | Discontinue bevacizumab |
| Hemorrhage (CNS or pulmonary) | Grade 2-4 | Discontinue bevacizumab |

| Event | CTCAE.v4.0 Grade | Action To Be Taken |
|---|---|---|
| Hemorrhage (non-CNS;<br>non-pulmonary) | Grade 3 | Patients receiving full-dose anticoagulation should discontinue bevacizumab For patients not on full-dose anticoagulation, hold bevacizumab until ALL of the following criteria are met: |
| | Grade 4 | Discontinue bevacizumab |
| RPLS (reversible posterior leu syndrome or PRES (posterior encephalopathy syndrome) | reversible | Hold bevacizumab in patients with symptoms/signs suggestive of RPLS; subsequent management should include MRI scans and control of HTN Discontinue bevacizumab upon diagnosis of RPLS |
| Wound dehiscence requiring intervention | medical or surgical | Discontinue bevacizumab |
| GI perforation, GI leak or fist | ula | Discontinue bevacizumab |
| Bowel obstruction | Grade 2 requiring medical intervention Grade 3-4 | <ul> <li>Hold bevacizumab until complete resolution, with a minimum of 4 weeks after surgery.</li> <li>Hold bevacizumab until complete resolution</li> <li>If surgery is required, patient may restart bevacizumab after full recovery from surgery, and at investigator's discretion</li> </ul> |
| Other unspecified bevacizumab-related AEs (except controlled nausea/vomiting). | Grade 3<br>Grade 4 | <ul> <li>Hold bevacizumab until symptoms resolve to ≤ grade 1</li> <li>Discontinue bevacizumab</li> <li>Upon consultation with the study chair, resumption of bevacizumab may be considered if a patient is benefiting from therapy and the grade 4 toxicity is transient, has recovered to ≤ grade 1 and unlikely to recur with retreatment</li> </ul> |

#### **7.4 Modality Review** (11/20/13)

The Medical Oncology Co-Chair, Jeffrey Raizer, M.D., will perform a Chemotherapy Assurance Review of all patients who receive or are to receive chemotherapy in this trial. The goal of the review is to evaluate protocol compliance. The review process is contingent on timely submission of chemotherapy treatment data as specified in <a href="Section 12.1">Section 12.1</a>. The scoring mechanism is: Per Protocol/Acceptable Variation, Not Per Protocol, and Not Evaluable. A report is sent to each institution once per year to notify the institution about compliance for each case reviewed in that year.

The Medical Oncology Co-Chair, Jeffrey Raizer, M.D., will perform a Quality Assurance Review after complete data for the first 20 cases enrolled has been received at NRG Oncology. Dr. Raizer will perform the next review after complete data for the next 20 cases enrolled has been received at NRG Oncology. The final cases will be reviewed within 3 months after this study has reached the target accrual or as soon as complete data for all cases enrolled has been received at NRG Oncology, whichever occurs first.

#### **7.5** Adverse Events (2/27/14)

This study will utilize the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 for adverse event (AE) reporting. The CTCAE version 4.0 is located on the CTEP website at http://ctep.cancer.gov/protocolDevelopment/electronic\_applications/ctc.htm. All appropriate treatment areas should have access to a copy of the CTCAE version 4.0.

Adverse events (AEs) that meet expedited reporting criteria defined in the table(s) below will be reported via the CTEP-AERS (CTEP Adverse Event Reporting System) application accessed via either the CTEP web site (<a href="https://eapps-ctep.nci.nih.gov/ctepaers/pages/task?rand=1390853489613">https://eapps-ctep.nci.nih.gov/ctepaers/pages/task?rand=1390853489613</a>).

#### 7.5.1 Adverse Events (AEs)

**Definition of an AE**: Any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. Therefore, an AE can be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not considered related to the medicinal (investigational) product (attribution of unrelated, unlikely, possible, probable, or definite). (International Conference on Harmonisation [ICH], E2A, E6). [CTEP, NCI Guidelines: Adverse Event Reporting Requirements. February 29, 2012.

## 7.5.2 <u>Serious Adverse Even</u>ts (SAEs)

Serious adverse events (SAEs) that meet expedited reporting criteria defined in the table in <a href="Section 7.6">Section 7.6</a> will be reported via CTEP-AERS. SAEs that require 24 hour CTEP-AERS notification are defined in the expedited reporting table in <a href="Section 7.6">Section 7.6</a>. Contact the CTEP-AERS Help Desk if assistance is required.

**Definition of an SAE**: Any adverse drug event (experience) occurring at any dose that results in any of the following outcomes:

- Death:
- A life-threatening adverse drug experience;
- Inpatient hospitalization or prolongation of existing hospitalization;
- A persistent or significant disability/incapacity;
- A congenital anomaly/birth defect;
- Important medical events that may not result in death, be life threatening, or require
  hospitalization may be considered an SAE, when, based upon medical judgment, they
  may jeopardize the patient and may require medical or surgical intervention to prevent
  one of the outcomes listed in the definition.

Due to the risk of intrauterine exposure of a fetus to potentially teratogenic agents, the pregnancy of a study participant must be reported via CTEP-AERS in an expedited manner.

#### 7.5.3 Acute Myeloid Leukemia (AML) or Myelodysplastic Syndrome (MDS)

AML or MDS that is diagnosed as a secondary malignancy during or subsequent to treatment in patients on NCI/CTEP-sponsored clinical trials must be reported via the CTEP-AERS within 30 days of AML/MDS diagnosis.

#### Secondary Malignancy

A secondary malignancy is a cancer caused by treatment for a previous malignancy (e.g., treatment with investigational agent/intervention, radiation or chemotherapy). A secondary malignancy is not considered a metastasis of the initial neoplasm.

CTEP requires all secondary malignancies that occur following treatment with an agent under an NCI IND/IDE be reported via CTEP-AERS. Three options are available to describe the event:

- Leukemia secondary to oncology chemotherapy (e.g., acute myelocytic leukemia [AML])
- Myelodysplastic syndrome (MDS)
- Treatment-related secondary malignancy
Any malignancy possibly related to cancer treatment (including AML/MDS) should also be reported via the routine reporting mechanisms outlined in each protocol.

#### Second Malignancy

A second malignancy is one unrelated to the treatment of a prior malignancy (and is NOT a metastasis from the initial malignancy). Second malignancies require ONLY routine reporting via CDUS unless otherwise specified.

#### 7.6 CTEP-AERS Expedited Reporting Requirements (2/27/14)

All serious adverse events that meet expedited reporting criteria defined in the reporting table below will be reported via CTEP-AERS, the CTEP Adverse Event Reporting System, accessed via the CTEP web site, <a href="https://eapps-ctep.nci.nih.gov/ctepaers/pages/task?rand=1390853489613">https://eapps-ctep.nci.nih.gov/ctepaers/pages/task?rand=1390853489613</a>.

Submitting a report via CTEP-AERS serves as notification to NRG Oncology and satisfies NRG Oncology requirements for expedited adverse event reporting.

CTEP-AERS provides a radiation therapy-only pathway for events experienced that involve radiation therapy only. These events must be reported via the CTEP-AERS radiation therapy-only pathway.

In the rare event when Internet connectivity is disrupted, a 24-hour notification must be made to the NRG Oncology Office at 1-800-227-5463, ext. 4189, for instances when Internet fails. Once internet connectivity is restored, an AE report submitted by phone must be entered electronically into CTEP-AERS.

- CTEP-AERS-24 Hour Notification requires that a CTEP-AERS 24-hour notification is
  electronically submitted within 24 hours of learning of the adverse event. Each CTEP-AERS
  24-hour notification must be followed by a CTEP-AERS 5 Calendar Day Report. Serious
  adverse events that require 24 hour CTEP-AERS notification are defined in the expedited
  reporting table below.
- Supporting source document is not mandatory. However, if the CTEP-AERS report indicates
  in the Additional Information section that source documentation will be provided, then it is
  expected. If supporting source documentation accompanies a CTEP-AERS report, include
  the protocol number, patient ID number, and CTEP-AERS ticket number on each page, and
  fax supporting documentation to the NRG Oncology dedicated SAE FAX, 215-717-0990.
- A serious adverse event that meets expedited reporting criteria outlined in the following table
  but is assessed by the CTEP-AERS as "expedited reporting NOT required" must still be
  reported to fulfill NRG Oncology safety reporting obligations. Sites must bypass the "NOT
  Required" assessment; the CTEP-AERS allows submission of all reports regardless of the
  results of the assessment.

CTEP defines expedited AE reporting requirements for phase 2 and 3 trials as described in the table below. **Important:** All AEs reported via CTEP-AERS also must be reported on the AE section of the appropriate case report form (see <u>Section 12.1</u>).

Late Phase 2 and Phase 3 Studies: Expedited Reporting Requirements for Adverse Events that Occur on Studies under an IND/IDE within 30 Days of the Last Administration of the Investigational Agent/Intervention <sup>1, 2</sup>

#### FDA REPORTING REQUIREMENTS FOR SERIOUS ADVERSE EVENTS (21 CFR Part 312)

**NOTE:** Investigators <u>MUST</u> immediately report to the sponsor (NCI) <u>ANY</u> Serious Adverse Events, whether or not they are considered related to the investigational agent(s)/intervention (21 CFR 312.64)

An adverse event is considered serious if it results in **ANY** of the following outcomes:

- 1) Death
- 2) A life-threatening adverse event
- 3) An adverse event that results in inpatient hospitalization or prolongation of existing hospitalization for ≥ 24 hours
- A persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions
- 5) A congenital anomaly/birth defect.
- 6) Important Medical Events (IME) that may not result in death, be life threatening, or require hospitalization may be considered serious when, based upon medical judgment, they may jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the outcomes listed in this definition. (FDA, 21 CFR 312.32; ICH E2A and ICH E6).

<u>ALL SERIOUS</u> adverse events that meet the above criteria <u>MUST</u> be immediately reported to the NCI via CTEP-AERS within the timeframes detailed in the table below.

| Hospitaliz-<br>ation | Grade 1<br>Timeframes | Grade 2<br>Timeframes | Grade 3<br>Timeframes | Grade 4 & 5<br>Timeframes |
|---|---|---|---|---|
| Resulting in Hospitalization ≥ 24 hrs | 10 Calendar Days | | 24-Hour 5 Calendar | |
| Not resulting in<br>Hospitalization<br>≥ 24 hrs | Not required 10 Calend | | 10 Calendar Days | Days |

**NOTE**: Protocol specific exceptions to expedited reporting of serious adverse events are found in the Specific Protocol Exceptions to Expedited Reporting (SPEER) portion of the CAEPR

#### **Expedited AE reporting timelines are defined as:**

- "24-Hour; 5 Calendar Days" The AE must initially be reported via CTEP-AERS within 24 hours of learning of the AE, followed by a complete expedited report within 5 calendar days of the initial 24-hour report.
- "10 Calendar Days" A complete expedited report on the AE must be submitted within 10 calendar days of learning of the AE.

<sup>1</sup>Serious adverse events that occur more than 30 days after the last administration of investigational agent/intervention and have an attribution of possible, probable, or definite require reporting as follows:

#### Expedited 24-hour notification followed by complete report within 5 calendar days for:

All Grade 4, and Grade 5 AEs

#### Expedited 10 calendar day reports for:

- Grade 2 adverse events resulting in hospitalization or prolongation of hospitalization
- Grade 3 adverse events

Date: May 5, 2011

<sup>&</sup>lt;sup>2</sup> For studies using PET or SPECT IND agents, the AE reporting period is limited to 10 radioactive half lives, rounded UP to the nearest whole day, after the agent/intervention was last administered. Footnote "1" above applies after this reporting period.

# Additional Instructions or Exceptions to CTEP-AERS Expedited Reporting Requirements for Phase 2 and 3 Trials Utilizing an Agent under a CTEP-IND [or Non-CTEP IND]:

Not applicable.

#### 8.0 SURGERY

Not applicable to this study.

#### 9.0 OTHER THERAPY

#### 9.1 Permitted Supportive Therapy

All supportive therapy for optimal medical care will be given during the study period at the discretion of the attending physician(s) within the parameters of the protocol and documented on each site's source documents as concomitant medication.

- **9.1.1** Anticonvulsants: No limitations in type of anti-convulsants used.
- **9.1.2** Antiemetics: Prophylactic medications are not needed. For nausea, anti-emetics may be used based on the treating physician's preference.
- **9.1.3** Anticoagulants: These may be used for the treatment of DVT's or PE's if they occur. Preference should be given for LMW Heparins, but Coumadin is allowed.
- **9.1.4** Antidiarrheals: Used as needed per treating physician's discretion.
- **9.1.5** Analgesics: Used as needed per treating physician's discretion.
- **9.1.6** Hematopoietic Growth Factors: Used as needed per treating physician's discretion.
- **9.1.7** Herbal products: Are allowed but patients should inform treating physician and these should be recorded.
- **9.1.8** Nutritional supplementation: Are allowed but patients should inform treating physician and these should be recorded.

#### 9.2 Non-permitted Supportive Therapy

**9.2.1** Patients should avoid the use of medications that have anti-oxidant properties during radiation.

#### 10.0 TISSUE/SPECIMEN SUBMISSION

NOTE: Patients must be offered the opportunity to participate in the correlative components of the study, such as tissue/specimen submission or quality of life assessment. If the patient consents to participate in the tissue/specimen component of the study, the site is required to submit the patient's specimens as specified in <a href="Section 10.0">Section 10.0</a> of the protocol. Sites are <a href="not">not</a> permitted to delete the tissue/specimen component from the protocol or from the sample consent.

#### 10.1 Tissue/Specimen Submission

The NRG Oncology Biospecimen Bank at the University of California San Francisco acquires and maintains high quality specimens from NRG Oncology trials. Tissue from each block is preserved through careful block storage and processing. NRG Oncology encourages participants in protocol studies to consent to the banking of their tissue. The NRG Oncology Biospecimen Bank provides tissue specimens to investigators for translational research studies. Translational research studies integrate the newest research findings into current protocols to investigate important biologic questions.

In this study, tissue will be submitted to the NRG Oncology Biospecimen Bank for the purpose of tissue banking and translational research (highly recommended).

# 10.2 Specimen Collection for Banking and Translational Research (Highly Recommended) (10/9/14)

For patients who have consented to participate in the specimen collection component of the study.

The following must be provided in order for the case to be evaluable for the NRG Oncology Biospecimen Bank:

- **10.2.1** <u>Tissue</u> (For collection, processing and shipping information please see Specimen Collection Summary below and Appendix III.)
  - One H&E stained slide (slide can be a duplicate cut stained H&E of the diagnostic slide (block); it does not have to be the diagnostic slide itself)
  - A corresponding paraffin-embedded tissue block of the tumor (the block must match the H&E being submitted) or a 2 mm diameter core of tumor tissue, punched from the tissue block containing the tumor with a punch tool and submitted in a plastic tube labeled with the surgical pathology number. <u>Note</u>: A kit with the punch, tube, and instructions can be obtained free of charge from the NRG Oncology Biospecimen Bank. Block or core must be clearly labeled with the pathology identification number and block number that corresponds to the Pathology Report (see below).
    - The submitted material must be from malignant tumor, not necrotic or fibrotic tissue. If the submitted material is reviewed and is not tumor, the site may be assessed a protocol violation.
  - A Pathology Report documenting that the submitted block or core contains tumor. The report
    must include the NRG Oncology protocol number and patient's case number. The patient's
    name and/or other identifying information should be removed from the report. The surgical
    pathology numbers and information must NOT be removed from the report.
  - A Specimen Transmittal (ST) Form clearly stating that tissue is being submitted for NRG Oncology Biospecimen Bank; if for translational research, this should be stated on the form.
     The form must include the NRG Oncology protocol number and patient's case number.
- **10.2.2** <u>Blood and Urine</u> (For collection, processing and shipping information please see Specimen Collection Summary below and <u>Appendix III</u>.)

A Specimen Transmittal Form documenting the type of Biospecimen, the date of collection of the biospecimen; the NRG Oncology protocol number, the patient's case number, time point of study, and method of storage, for example, stored at -80° C, must be included.

#### 10.2.3 Storage Conditions for All Specimens

Store frozen specimens at -80° C (-70°C to -90°C) until ready to ship. If a -80°C Freezer is not available:

• Samples can be stored short term in a -20° C freezer (non-frost free preferred) for up to one week (please ship out Monday-Wednesday only; Canada: Monday-Tuesday).

#### <u>OR</u>

• Samples can be stored in plenty of dry ice for up to one week, replenishing daily (ship out Monday-Wednesday only; Canada: Monday-Tuesday).

#### OR:

• Samples can be stored in liquid nitrogen vapor phase (ship out Monday-Wednesday only; Canada: Monday-Tuesday).

Please indicate on the ST Form the storage conditions used and time stored.

#### 10.2.4 Specimen Collection Summary

| Specimens for Banking/Translational Research | | | |
|---|---|---|---|
| Specimens taken from patient: | Collected when: | Submitted as: | Shipped: |
| Representative H&E stained slides of the primary tumor | Pre-treatment | H&E stained slide | Slide shipped ambient |
| A paraffin-embedded tissue block of the primary tumor taken before initiation of treatment or a 2 mm diameter core of tissue, punched from the tissue block with a punch tool | Pre-treatment | Paraffin-embedded<br>tissue block or punch<br>biopsy (must match the<br>H&E slide being<br>submitted) | Block or punch shipped<br>ambient. Cold packs are<br>recommended during<br>warm weather to help<br>prevent blocks from<br>melting |
| SERUM: 5-10 mL of whole blood in 1 red-top tube and centrifuge | <ul><li>(1) Pre-treatment</li><li>(2) 8 weeks after treatment initiation</li></ul> | Frozen serum samples containing 0.5 mL per aliquot in 1 mL cryovials (five to eight) | Serum sent frozen on dry ice via overnight carrier |
| PLASMA: 5-10 mL of<br>anticoagulated whole blood<br>in EDTA tube #1 (purple/<br>lavender top) and<br>centrifuge | <ul><li>(1) Pre-treatment</li><li>(2) 8 weeks after treatment initiation</li></ul> | Frozen plasma samples<br>containing 0.5 mL per<br>aliquot in 1 mL cryovials<br>(five to eight) | Plasma sent frozen on dry ice via overnight carrier |
| Whole blood for DNA: 5-10 mL of anticoagulated whole blood in EDTA tube #2 (purple/ lavender top) and mix | (1) Pre-treatment<br>(Note: if site missed this<br>timepoint they may collect<br>whole blood at any<br>timepoint or follow up visit,<br>but this must be noted on<br>the ST Form) | Frozen whole blood<br>samples containing 1.0<br>mL per aliquot in 1 mL<br>cryovials (three-five) | Whole blood sent frozen on dry ice via overnight carrier |
| 10-20 mL clean-catch urine | (1) Pre-treatment (2) 8 weeks after treatment initiation | Two 5-10 mL urine aliquots in 2 sterile 15 ml polypropylene centrifuge tubes. Store frozen at -20° or 80° C | Urine sent frozen on dry ice via overnight carrier |

#### **10.2.5** Submit materials for Specimen Banking, Translational Research as follows:

U. S. Postal Service Mailing Address: <u>For Non-frozen Specimens Only</u> NRG Oncology Biospecimen Bank University of California San Francisco UCSF Box 1800 2340 Sutter Street, Room S341 San Francisco, CA 94143-1800

Courier Address (FedEx, UPS, etc.): <u>For Trackable FFPE and ALL Frozen Specimens</u>

NRG Oncology Biospecimen Bank
University of California San Francisco

2340 Sutter Street, Room S341 San Francisco, CA 94115

Questions: 415-476-7864/FAX 415-476-5271; RTOG@ucsf.edu

#### **10.3** Reimbursement (4/15/14)

Please note that with the start of the new NCI National Clinical Trials Network (NCTN) Program, NCI funds for reimbursement for protocol-specified biospecimen materials will be distributed per

the requirements/methods specified by the new NCTN Program. This information will be made available with the other registration materials in the Oncology Patient Enrollment Network (OPEN) portal system. OPEN will serve as the registration system for all patient enrollments onto NCI-sponsored NCTN trials, including this study, which will be transitioned into the new Program from the NCI-sponsored Cooperative Group Clinical Trials Program.

#### 10.4 Confidentiality/Storage

(See the Patient Tissue Consent Frequently Asked Questions, <a href="http://www.rtog.org/Researchers/BiospecimenResource/BiospecimenResourceFAQs.aspx">http://www.rtog.org/Researchers/BiospecimenResource/BiospecimenResourceFAQs.aspx</a> for further details.)

- **10.4.1** Upon receipt, the specimen is labeled with the NRG Oncology protocol number and the patient's case number only. The NRG Oncology Biospecimen Bank database only includes the following information: the number of specimens received, the date the specimens were received, documentation of material sent to a qualified investigator, type of material sent, and the date the specimens were sent to the investigator. No clinical information is kept in the database.
- **10.4.2** Specimens for tissue banking will be stored for an indefinite period of time. Specimens for the translational research component of this protocol will be retained until the study is terminated, unless the patient has consented to storage for future studies. If at any time the patient withdraws consent to store and use specimens, the material will be returned to the institution that submitted it.

#### 11.0 PATIENT ASSESSMENTS

- 11.1 Study Parameters: See Appendix I. See below for additional details. (11/20/13)
- **11.1.1** Urine should be assessed via dipstick or random urine creatinine and protein before each dose of bevacizumab. If dipstick is > 2 + then a UPC ratio should be performed.
- **11.1.2** Vital signs should be assessed before each dose of bevacizumab (on treatment day) to make sure there is no increase in blood pressure.
- **11.1.3** MR diffusion and perfusion imaging at 8 and 24 weeks post-treatment start is optional but strongly recommended. Repeat MR diffusion and perfusion imaging at progression is optional but strongly recommended as further confirmation of true tumor progression and not radiation necrosis.

#### 11.2 Measurement of Response

The primary measure of response will be by serial measures of the product of the two largest cross-sectional diameters using MacDonald Criteria. Response will also be evaluated in this study using the international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee [JNCI 92(3): 205-216, 2000], see Section 11.4.

#### 11.2.1 Complete Response (CR)

Requires all of the following: complete disappearance of the measurable enhancing lesion sustained for at least 4 weeks; no new lesions; and no corticosteroids.

#### **11.2.2** Partial Response (PR)

Requires all of the following: ≥ 50% decrease compared with baseline in the sum of products of perpendicular diameters of the measurable enhancing lesion sustained for at least 4 weeks; no new lesions; and stable or reduced corticosteroid dose.

#### 11.2.3 Stable Disease (SD)

Requires all of the following: does not qualify for complete response, partial response, or progression and is receiving stable or decreasing doses of steroids. This will not require a confirmatory scan.

#### **11.2.4** Progression (P)

Defined by any of the following: ≥ 25% increase in sum of the products of perpendicular diameters of enhancing lesions provided that the patient has not had his/her dose of steroids decreased since the last evaluation period; and any new lesions. This will not require a confirmatory scan. A concomitant decrease in steroid dose will rule out a progression designation during the initial 12 weeks after completion of RT.

#### **11.2.5** Pseudo-progression

Due to possible radiation effects using large dose per fraction, the initial scan 6 weeks following RT should NOT be used to declare progression. In the absence of neurologic worsening OR a new distant area of tumor, the initial post-radiation scan should not be used to declare progression. Progressive worsening on subsequent imaging studies usually distinguishes true progression from pseudo-progression.

11.2.6 If true progression is determined by subsequent imaging, then the date of progression returns to the earlier date with increasing mass.

#### 11.3 **Criteria for Evaluation of Therapy Effectiveness**

- 11.3.1 Tumor response and regrowth can frequently be difficult to measure directly. Serial neurological exams and CT/MRI scans may provide a guide to the actual course. Time interval to progression will be measured from registration until deterioration is documented by the individual investigator using these guides. The patient should consistently be followed with the same diagnostic imaging study (CT or MRI). (NOTE: CT option ONLY for patients unable to undergo MR imaging because of non-compatible devices.)
- 11.3.2 Overall survival will be measured from registration until death. Progression-free survival will be measured from registration until the first occurrence of progression or death.
- 11.3.3 The quality of survival will be measured by neurological functional classification and performance
- **11.3.4** Toxicities will be measured using the CTCAE criteria, version 4.0.

#### 11.4 **RANO Response Criteria**

Efficacy determinations using RANO response criteria (Wen 2010) also will be obtained.

#### 11.4.1 Response Criteria

Radiographic response should be determined in comparison to the tumor measurement obtained at pretreatment baseline for determination of response, and the smallest tumor measurement at either pretreatment baseline or following initiation of therapy for determination of progression. The tables below outline the criteria for radiographic changes following therapy and summarize RANO response criteria. In the event that the radiographic changes are equivocal and it is unclear whether the patient is stable or has developed progressive disease, it is permissible to continue treatment and observe the patient closely, for example at 4 weekly intervals. If subsequent imaging studies demonstrate that progression has occurred, the date of progression should be the scan at which this issue was first raised.

All measurable and non-measurable lesions should be assessed using the same techniques as baseline. Ideally patients should be imaged on the same MRI, or least with the same magnet strength, for the duration of the study to reduce difficulties in interpreting changes.

All measurable and non-measurable lesions must be assessed using the same techniques as baseline.

43

#### Criteria for Response Assessment Incorporating MRI and Clinical Factors

#### **Complete Response:**

Requires all of the following:

- a) Complete disappearance of all enhancing measurable and non-measurable disease sustained for at least 4 weeks.
- b) No new lesions.
- c) Stable or improved non-enhancing (T2/FLAIR) lesions.
- d) Patients must be off corticosteroids (or on physiologic replacement doses only).
- e) Stable or improved clinically.

Note: Patients with non-measurable disease only cannot have a complete response. The best response possible is stable disease.

#### Partial Response:

Requires all of the following:

- a) Greater than or equal to 50% decrease compared to baseline in the sum of products of perpendicular diameters of all measurable enhancing lesions sustained for at least 4 weeks.
- b) No progression of non-measurable disease.
- c) No new lesions.
- d) Stable or improved non-enhancing (T2/FLAIR) lesions on same or lower dose of corticosteroids compared to baseline scan.
- e) The corticosteroid dose at the time of the scan evaluation should be no greater than the dose at time of baseline scan.
- f) Stable or improved clinically.

Note: Patients with non-measurable disease only cannot have a partial response. The best response possible is stable disease.

#### Stable Disease:

Requires all of the following:

- a) Does not qualify for complete response, partial response, or progression.
- b) Stable non-enhancing (T2/FLAIR) lesions on same or lower dose of corticosteroids compared to baseline scan. In the event that the corticosteroid dose was increased for new symptoms and signs without confirmation of disease progression on neuroimaging, and subsequent follow-up imaging shows that this increase in corticosteroids was required because of disease progression, the last scan considered to show stable disease will be the scan obtained when the corticosteroid dose was equivalent to the baseline dose.
- c) Stable clinically.

#### **Progression:**

Defined by any of the following:

- a) Greater than > 25% increase in sum of the products of perpendicular diameters of enhancing lesions compared to the smallest tumor measurement obtained either at baseline (if no decrease) or best response, on stable or increasing doses of corticosteroids.\*
- b) Significant increase in T2/FLAIR non-enhancing lesion on stable or increasing doses of corticosteroids compared to baseline scan or best response following initiation of therapy,\* not due to co-morbid events (e.g. radiation therapy, demyelination, ischemic injury, infection, seizures, post-operative changes, or other treatment effects).
- c) Any new lesion.
- d) Clear clinical deterioration not attributable to other causes apart from the tumor (e.g. seizures, medication side effects, complications of therapy, cerebrovascular events, infection, etc.) or changes in corticosteroid dose.
- e) Failure to return for evaluation due to death or deteriorating condition.
- f) Clear progression of non-measurable disease.
- \*Stable doses of corticosteroids include patients not on corticosteroids

**Summary of RANO Response Criteria** 

| Summary of the troopened striction | | | | |
|---|---|---|---|---|
| <u>Criterion</u> | <u>CR</u> | <u>PR</u> | <u>SD</u> | <u>PD</u> # |
| T1-Gd + | None | ≥ 50% ↓ | < 50% ↓ - < 25% ↑ | ≥ 25% ↑* |
| T2/FLAIR | Stable or ↓ | Stable or ↓ | Stable or ↓ | <b>^</b> * |
| New Lesion | None | None | None | Present* |
| Corticosteroids | None | Stable or ↓ | Stable or ↓ | NA** |
| Clinical Status | Stable or ↑ | Stable or ↑ | Stable or ↑ | <b>↓</b> * |
| Requirement for response | All | all | All | Any* |

Abbreviations: RANO, Response Assessment in Neuro-Oncology; CR=complete response; PR=partial response; SD=stable disease; PD=progressive disease; FLAIR, fluid-attenuated inversion recovery; ↓ = decrease: ↑ = increase

NA\*\*: Increase in corticosteroids alone will not be taken into account in determining progression in the absence of persistent clinical deterioration.

#### **11.4.2** Efficacy Assessments

- <u>Progression free survival (PFS)</u> will be defined from the time the patient enters the study until there is clinical or radiographic evidence of progressive disease (see definition of PD above).
- <u>Overall survival (OS)</u> will be defined from the time the patient enters the study to the date of death. Patients not known to have died will be censored for survival as of the last date known alive.
- PFS and overall survival will be estimated by using the Kaplan-Meier method.
- The primary endpoint for this study is overall survival.

#### 11.5 Criteria for Discontinuation of Protocol Treatment

- Progression of disease (See Section 11.2)
- Unacceptable toxicity to the patient (at the discretion of the treating physician) Reasons for removal must be clearly documented on the appropriate case report form/flow sheet, and NRG Oncology data management must be notified.

If protocol treatment is discontinued, follow up and data collection will continue as specified in the protocol.

<sup>\*</sup> Progression occurs when any of the criteria with \* is present.

#### 12.0 DATA COLLECTION

Data should be submitted to:

# NRG Oncology\* 1818 Market Street, Suite 1600 Philadelphia, PA 19103

#### \*If a data form is available for web entry, it must be submitted electronically.

Patients will be identified by initials only (first middle last); if there is no middle initial, a hyphen will be used (first-last). Last names with apostrophes will be identified by the first letter of the last name.

#### **12.1** Summary of Data Submission (10/9/14)

report to NRG Oncology

Pathology Report (P1) to mail a copy of the

ItemDueDemographic Form (A5)Within 2 weeks after registrationInitial Evaluation Form (I1)

Treatment Form (**TF**) At completion of each 8-week period (4 doses of

bevacizumab per TF form if no protocol

modification)

Follow-up Form (F1)

At the time of progression and at death. AFTER

progression or treatment discontinuation: every 2 months for 1 year, then every 6 months for 1

year, then annually.

MRI scans and Reports (MR, ME) Pre-study (complete series) (see Section 12.2)

Progression to TRIAD (see Section 12.2)

**12.2 Summary of Dosimetry Digital Data Submission** (Submit to TRIAD; see Section 5.5 for account access and installation instructions) (4/15/14)

#### **Preliminary Dosimetry Information**

Digital Data Submission - Treatment

Within 1 week of start of RT

Digital data submission includes the following, all in DICOM format:

- CT data, critical normal structures, all GTV, CTV, and PTV contours
- Digital beam geometry beam sets
- Single dose file for concurrently treated beams
- Digital DVH data for all required critical normal structures, GTV, CTV, and PTVs for total dose plan
- All required structures **MUST** be labeled per Table in Section 6.5.1.

 The "RTOG 1205 Datasheet" is available in the Forms section of the of the NRG Oncology/RTOG web site, <a href="http://www.rtog.org/ClinicalTrials/ProtocolTable/StudyDetails.aspx?study=1">http://www.rtog.org/ClinicalTrials/ProtocolTable/StudyDetails.aspx?study=1</a>
 205. Submit via TRIAD with the digital data listed above.

Upon submission of any digital data via TRIAD, complete an online digital data submission form (DDSI) located on the NRG Oncology/RTOG web site at http://www.rtog.org/ClinicalTrials/ProtocolTable/StudyDetails.aspx?study=1205

<u>Item</u> <u>Due</u>

**MRI SUBMISSION** 

Pre-study MRI (the Scan used to delineate the target volumes for planning. Submit the entire series via TRIAD

Final Dosimetry Information
Radiotherapy Form (T1) via the web
Daily Treatment Record (T5) on paper to HQ

Within 1 week of RT end

**NOTE:** ALL SIMULATION AND PORTAL FILMS AND/OR DIGITAL FILM IMAGES WILL BE KEPT BY THE INSTITUTION AND ONLY SUBMITTED IF REQUESTED.

#### 13.0 STATISTICAL CONSIDERATIONS

**13.1** Study Endpoints (11/20/13)

#### **13.1.1** Primary Endpoint

Overall Survival, defined as the interval from randomization to death due to any cause.

#### **13.1.2** Secondary Endpoints

- Objective response
- 6-month progression-free survival
- Progression-free survival, defined as the interval from randomization to progression or death, whichever occurs first
- Treatment adverse events
- Grade 3+ acute or delayed CNS toxicity

#### 13.2 Sample Size and Power Justification

The primary objective of this study is to determine whether re-irradiation plus bevacizumab (experimental arm) will improve the overall survival compared to bevacizumab alone (control arm). The design will be a randomized phase II screening trial as proposed by Rubinstein et al (2005). The randomization of experimental and control arms is 1:1. The null hypothesis is that the overall survival for both arms is 9 months, based on data from RTOG 0625/ACRIN 6677 and the BRAIN study. The alternative hypothesis is that patients receiving IMRT plus bevacizumab will have an improvement in overall survival to 13 months, based on the Gutin data. With 160 eligible subjects, there will be 80% power to detect a 31% reduction in the hazard ratio to 0.69 at the significance level of 0.10 (one-sided). Analysis will be performed when 135 events (deaths) are reported, expected to occur 16 to 21 months after trial closure. Guarding against up to a 10% ineligibility rate, the final target accrual for this study will be 178 cases.

#### 13.3 Patient Accrual

Based on the monthly accrual for a prior RTOG recurrent glioblastoma phase II study (RTOG 0625), this study is projected to accrue 10 cases/month. Therefore, the target accrual should be completed within 22 months of study activation, allowing slow accrual in the first 6 months. If the average monthly accrual (6 months after trial activation) is less than 5 patients, the study will be re-evaluated with respect to feasibility.

#### **13.4** Patient Stratification and Randomization (4/15/14)

A randomized phase II trial will be conducted for bevacizumab-naïve recurrent GBM patients. Age and Karnofsky performance status (KPS) are demonstrated to be prognostic of survival for recurrent GBM (Carson 2007). In addition, previous RTOG recurrent GBM trials (RTOG 0625, 0627) show that age, KPS, and resection type have prognostic value in overall survival. Therefore, for this NRG Oncology recurrent GBM study, patients will be stratified by age (<50 vs. ≥50), KPS (60 vs. 70-80 vs.90-100), and resection type (yes vs. no/biopsy only), and then randomized to either the control arm or experimental arm in a permuted block design using the method described by Zelen (1974).

#### 13.5 Analyses Plans

#### **13.5.1** Statistical Methods

Overall and progression-free survival rates will be estimated using the Kaplan-Meier method (Kaplan 1958), and differences between treatment arms will be tested in the log-rank test (Mantel 1966). Overall survival will be measured from the date of randomization to the date of death or, otherwise, the last follow-up date on which the patient was reported alive. Progression-free survival will be measured from the date of randomization to the date of first progression or death or, otherwise, the last follow-up date on which the patient was reported alive.

Objective response rate, grade 3+ toxicities rate, acute or delayed CNS toxicity rate, and 6-month progression-free survival rate, will be estimated using an exact binomial distribution together with 95% confidence interval. The difference between the 2 groups will be tested using a chi square test. In terms of grade 3+ toxicity and acute/delayed toxicity, all patients receiving any protocol treatment (bevacizumab or combination of RT with bevacizumab) should be included. For the statistical comparison of the primary endpoint (overall survival), the type I error is set as 0.1 (1-sided), while for all the secondary endpoints, the statistical comparison between groups will serve as an exploratory purpose without multiple comparison adjustment, with type I error of 0.05 (2-sided) for each comparison.

Multivariate analyses with the Cox proportional hazard model (Cox 1972) for overall and progression-free survival will be performed with the stratification variables as fixed variables to assess the treatment effect adjusting patient-specific risk factors. The covariates evaluated for the multivariate models are assigned protocol treatment, tumor volume at the time of treatment, time since original diagnosis, stratification factors, and other prognostic factors. Proportional hazard assumptions will be checked using different graphical or time-varying coefficients testing methods. If the data clearly do not follow proportional hazards, other statistical models will be used to fit the data instead. Possible alternatives are to use the stratified Cox proportional hazard model, accelerated failure model, or partition the time axis into sections where proportional hazard assumption holds.

#### **13.5.2** Interim Toxicity and Futility Analysis

Due to a possible increased incidence of grade 3+ CNS toxicity (possibly, probably, or definitely related to treatment) occurring during the first 6 months post RT in the experimental arm, a special interim analysis will be performed after the first 20 patients enrolled to the experimental arm have a minimum 6-month follow-up. If the incidence of grade 3+ CNS toxicity (based on RTOG 0625) is 20% higher, or 30%, in the experimental arm, the trial will be halted due to lack of safety. The interim toxicity analysis results will be reported to the NRG Oncology DMC. The DMC will then make a recommendation about the trial to the NRG Oncology Group Co-Chairs.

The interim futility analysis will be performed when 50% of the required events (68 deaths) are reported. The analysis will be performed on an intent-to-treat basis, with all eligible cases included in the treatment arm to which they were randomized regardless of what treatment the patients actually received. The primary endpoint, overall survival, will be tested. The futility will be tested using the conditional probability under the alterative hypothesis of detecting the hypothesized treatment benefit favoring the experimental arm at the final analysis given the observed data. The results from testing the treatment futility will be reported to the NRG Oncology DMC. The responsible statistician may recommend early reporting of the results and/or stopping

accrual (if applicable) of the trial if the conditional power is less than 0.1. The accrual rate, treatment compliance, safety of the treatments, and the importance of the study are also considered in making such a recommendation. The results will be reported to the RTOG DMC with the treatment blinded. The DMC will then make a recommendation about the trial to the NRG Oncology Group Co-Chair.

#### **13.5.3** Interim Analysis to Monitor Study Progress

Interim reports with statistical analyses are prepared every 6 months until the initial manuscript reporting the treatment results has been submitted. The reports contain:

- The patient accrual rate with a projected accrual completion date
- Accrual by institution
- The pretreatment characteristics of accrued patients
- The frequency and severity of toxicities
- The results of any completed study chair modality reviews

The interim reports will not contain the results from the treatment comparisons with respect to the efficacy endpoints (overall survival, progression-free survival, treatment response). The NRG Oncology DMC will review the accrual to the study and the rate of adverse events on the study at least twice per year until the initial results of the study have been presented to the scientific community.

#### **13.5.4** Significance Testing for Final Analysis

The final analysis will be performed on an intent-to-treat basis, such that all eligible cases on the study will be included in the arm to which they were randomized regardless of what treatment the patients actually received. The analysis to report the final results of treatment comparison between the experimental arm and the control arm will be undertaken when 135 events (deaths) have been reported. A one-sided log-rank test will be performed to test the difference in overall survival between the two treatment arms. If the p value is less than protocol-specified 0.10 (one sided), the study statistician will reject the null hypothesis and conclude that the experimental arm (re-radiation plus bevacizumab) is promising in prolonging overall survival, therefore supporting the development of a confirmatory phase III trial comparing this regimen to the current standard treatment. All information reported in the interim analyses to monitor the study progress (above) and the treatment compliance with respect to re-radiation and chemotherapy will also be included in the final report.

**13.5.5** This study will be monitored by the Clinical Data Update System (CDUS) version 3.0. Cumulative CDUS data will be submitted quarterly by electronic means. Reports are due January 31, April 30, July 31, and October 31.

#### 13.6 Gender and Minorities

In conformance with the National Institutes of Health (NIH) Revitalization Act of 1993 with regard to inclusion of women and minorities in clinical research, both men and women of all races and ethnic groups are eligible for this study. We will also analyze treatment differences by gender, race, and ethnicity. The following table lists the projected accrual for each racial and ethnic group based upon previous RTOG recurrent GBM trials.

**Projected Distribution of Gender and Minorities** 

| | | Gender | |
|----------------------------------------|---------|--------|-------|
| Ethnic Category | Females | Males | Total |
| Hispanic or Latino | 10 | 13 | 23 |
| Not Hispanic or Latino | 67 | 88 | 155 |
| Ethnic Category: Total of all subjects | 77 | 101 | 178 |
| | | Gender | |
| Racial Category | Females | Males | Total |
| American Indian or Alaskan Native | 1 | 1 | 2 |
| Asian | 3 | 3 | 6 |
| Black or African American | 6 | 6 | 12 |

| | | Gender | |
|-------------------------------------------|---------|--------|-------|
| Ethnic Category | Females | Males | Total |
| Native Hawaiian or other Pacific Islander | 1 | 1 | 2 |
| White | 66 | 90 | 156 |
| Racial Category: Total of all subjects | 77 | 101 | 178 |

#### **REFERENCES**

Brandes AA. State-of-the-art treatment of high-grade brain tumors. Semin Oncol. 2003;30:4-9.

Brenner DJ, Martel MK, Hall EJ. Fractionated regimens for stereotactic radiotherapy of recurrent tumors in the brain. *Int J Radiat Oncol Biol Phys.* 1997;21:819-824.

Carson KA, Grossman SA, Fisher JD, et al. Prognostic factors for survival in adult patients with recurrent glioma enrolled onto the new approaches to brain tumor therapy CNS consortium phase I and II clinical trials. *J Clin Oncol*. 2007;25:2601-2606.

Cho KH, Hall WA, Gerbi BJ, et al. Single dose versus fractionated stereotactic radiotherapy for recurrent high-grade gliomas. *Int J Radiat Oncol Biol Phys.* 1999;45:1133-1141.

Combs SE, Thilmann C, Edler L et al. Efficacy of fractionated stereotactic reirradiation in recurrent gliomas: Long-term results in 172 patients treated in a single institution. *J Clin Oncol*. 2005;23:8863-8869.

Cox DR. Regression models and life-tables. J Royal Statistical Society. 1972 (Series B);34:187-202.

Cuneo K, Vredenburgh J, Sampson JH et al, Safety and efficacy of stereotactic radiosurgery and adjuvant bevacizumab in patients with recurrent malignant gliomas, *Int J Radiat Oncol Biol Phys.* epub April 12, 2011.

Ellis LM, Hicklin DJ. VEGF-targeted therapy: mechanisms of anti-tumour activity. *Nat Rev Cancer*. 2008;8:579-591.

Fogh SE, Andrews DW, Glass J, et al. Hypofractionated stereotactic radiation therapy: an effective therapy for recurrent high-grade gliomas. *J Clin Oncol*. 2010;28:3048-3053.

Friedman HS, Prados M, Wen P, et al. Bevacizumab alone and in combination with irinotecan in recurrent glioblastoma. *J Clin Oncol.* 2009;27:4733-3740.

Gilbert MR, Wang M, Aldape K, et al. RTOG 0625: a phase II study of bevacizumab with irinotecan in recurrent glioblastoma. *J Clin Oncol*. 2009:27(15S):2011.

Gorski DH, Beckett MA, Jaskowiak NT, et al. Blockage of the vascular endothelial growth factor stress response increases the antitumor effects of ionizing radiation. *Cancer Res* 1999;59:3374-3378.

Grosu AL, Weber WA, Franz M, et al: Reirradiation of recurrent high-grade gliomas using amino acid PET (SPECT)/CT/MRI image fusion to determine gross tumor volume for stereotactic fractionated radiotherapy. *Int J Radiat Oncol Biol Phys.* 2005;63:511-519.

Gutin PH, Iwamoto FM, Beal K, et al. Safety and efficacy of bevacizumab with hypofractionated stereotactic irradiation for recurrent malignant gliomas. *Int J Radiat Oncol Biol Phys.* 2009;75:156-163.

Hasselbalch B, Lassen U, Hansen S, et al. Cetuximab, bevacizumab, and irinotecan for patients with primary glioblastoma and progression after radiation therapy and temozolomide: a phase II trial. *Neuro Oncol.* 2010;12:508-516.

Hovinga KE, Shimizu F, Wang R et al. Inhibition of notch signaling in glioblastoma targets cancer stem cells via an endothelial cell intermediate. *Stem Cells*. 2010;28:1019-1029.

Hudes RS, Corn BW, Werner-Wasik M, et al. A phase I dose escalation study of hypofractionated stereotactic radiotherapy as salvage therapy for persistent or recurrent malignant glioma. *Int J Radiat Oncol Biol Phys.*1999;43:293-298.

Jain RK, di Tomaso E, Duda DG, et al. Angiogenesis in brain tumours. *Nat Rev Neurosci*. 2007;8:610-622.

Kaplan EL, Meier P. Nonparametric estimation from incomplete observations. *J Am Stat Assoc.* 1958;53:457-481.

Kim HK, Thornton AF, Greenberg HS, et al. Results of re-irradiation of primary intracranial neoplasms with three-dimensional conformal therapy. *Am J Clin Oncol*.1997;20:358-363.

Kreisl TN, Kim L, Moore K, et al. Phase II trial of single-agent bevacizumab followed by bevacizumab plus irinotecan at tumor progression in recurrent glioblastoma. *J Clin Oncol.* 2009;27:4733-4740.

Laing RW, Warrington AP, Graham J, et al. Efficacy and toxicity of fractionated stereotactic radiotherapy in the treatment of recurrent gliomas (phase I/II study). *Radiother Oncol*. 1993;27:22-29.

Lai A, Tran A, Nghiemphu P, et al. Phase II study of bevacizumab plus temozolomide during and after radiation therapy for patients with newly diagnosed glioblastoma multiforme. *J Clin Oncol*. 2010;29:142-148.

Lederman G, Wronski M, Arbit E, et al. Treatment of recurrent glioblastoma multiforme using fractionated stereotactic radiosurgery and concurrent paclitaxel. *Am J Clin Oncol*. 2000;23:155-159.

Lee C-G, Heijn M, di Tomaso E, et al. Anti-vascular endothelial growth factor treatment augments tumor radiation response under normoxic or hypoxic conditions. *Cancer Res.* 2000;60:5565-5570

Levin VA, Bidaut L, Hou P, et al. Randomized double-blind placebo-controlled trial of bevacizumab therapy for radiation necrosis of the central nervous system. *Int J Radiat Oncol Biol Phys.* 2011;79:1487-1495.

Mantel N. Evaluation of survival data and two new rank order statistics arising in its consideration. *Cancer Chem Rep.* 1966;5:163-170.

Mayer R, Sminia P. Reirradiation tolerance of the human brain. *Int J Radiat Oncol Biol Phys.* 2008;70:1350-1360.

Nieder C, Astner ST, Mehta MP et al. Improvement, clinical course, and quality of life after palliative radiotherapy for recurrent glioblastoma. *Am J Clin Oncol*. 2008;31:300-305.

Niyazi M, Ganswindt U, Birgit S et al. Irradiation and bevacizumab in high-grade glioma retreatment settings. *Int J Radiat Oncol Biol Phys.* October 27, 2010. Epub ahead of print.

Provencio M, Sanchez A, Garrido P, et al. New molecular targeted therapies integrated with radiation therapy in lung cancer. *Clin Lung Cancer*. 2010;11:91-97.

Quant EC, Norden AD, Drappatz J, et al. Role of a second chemotherapy in recurrent malignant glioma patients who progress on bevacizumab. *Neuro Oncol.* 2009;11:550-555.

Reardon D, Desjardins A, Vredenburgh JJ, et al. Metronomic chemotherapy with daily, oral etoposide plus bevacizumab for recurrent malignant glioma: phase II study. *Br J Cancer*. 2009;101:1986-1994.

Rubinstein LV, Korn EL, Freidlin B, et al. Design issues of randomized phase II trials and a proposal for phase II screening trials. *J Clin Oncol*. 2005;23:7199-7206.

Sathornsumetee S, Desjardins A, Vredenburgh JJ, et al. Phase II study of bevacizumab and erlotinib in patients with recurrent malignant glioma. *Neuro Oncol.* 2010;12:1300-1310.

Stupp R, Mason WP, van den Bent MJ, et al. Radiotherapy plus concomitant and adjuvant temozolomide for glioblastoma. *New Engl J Med*. 2005;352:987-996.

VanderSpek L, Fisher B, Bauman G, et al. 3D conformal radiotherapy and cisplatin for recurrent malignant glioma. *Can J Neurol Sci.* 2008;35:57-64.

Verhoeff JJ, Lavini C, van Linde ME, et al. Bevacizumab and dose-intense temozolomide in recurrent high grade glioma. *Ann Oncol.* 2010;21:1723-1727.

Vredenburgh JJ, Desjardins A, Herndon JE, 2nd, et al. Phase II trial of bevacizumab and irinotecan in recurrent malignant glioma. *Clin Cancer Res.* 2007;13:1253-1259**a**.

Vredenburgh JJ, Desjardins A, Herndon JE, 2nd, et al. Bevacizumab plus irinotecan in recurrent glioblastoma multiforme. *J Clin Oncol.* 2007;25:4722-4729**b**.

Vredenburgh JJ, Cloughesy T, Samant M, et al, Corticosteroid use in patients with glioblastoma at first or second relapse treated with bevacizumab in the BRAIN study. *Oncologist*. 2010;15:1329-1334.

Vredenburgh JJ, Desjardins A, Reardon DA, et al. The addition of bevacizumab to standard radiation therapy and temozolomide followed by bevacizumab, temozolomide, and irinotecan for newly diagnosed glioblastoma. *Clin Cancer Res.* 2011:17:4119-4124.

Wong ET, Hess KR, Gleason MJ, et al. Outcomes and prognostic factors in recurrent glioma patients enrolled onto phase II clinical trials. *J Clin Oncol.* 1999;17:2572-2578.

Zelen M. (1974). The randomization and stratification of patients to clinical trials. *J Chronic Dis.* 27:365-75.

## **APPENDIX I: STUDY PARAMETER TABLES** (10/9/14)

## **Pre-Treatment Assessments**

| Assessment | Prior to registration | Within 14 days prior to registration | Pre-Treatment |
|---|---|---|---|
| Histopath dx | X | rogionanon | |
| (P1: pathology | ^ | | |
| report to be | | | |
| mailed to HQ per | | | |
| section 12.0) | | | |
| History | | X | |
| Physical | | X | |
| Neurological | | Х | |
| exam | | | |
| Tumor imaging | | Within 21 days | |
| MRI/CT scan (pts | | | |
| without recent | | | |
| resection; see | | | |
| Section 3.1.1for | | | |
| details) (MR | | | |
| diffusion and | | | |
| perfusion imaging | | | |
| strongly | | | |
| recommended) | | | |
| Tumor imaging | And recommended to be within | | |
| MRI/CT scan (pts | 96 h post-surgery | | |
| | 96 II post-surgery | | |
| with recent | | | |
| resection; see | | | |
| Section 3.1.4 for | | | |
| details) (MR | | | |
| diffusion and | | | |
| perfusion imaging | | | |
| strongly | | | |
| recommended) | | | |
| Karnofsky status | | X | |
| CBC w/ | | X | |
| differential | | | |
| Bilirubin | | X | |
| SGOT or AST | | | |
| Serum creatinine | | Х | |
| Urine protein: | | X<br>X | |
| creatinine or urine | | | |
| dipstick | | | |
| Serum pregnancy | | Within 7 days | |
| test (if applicable) | | vvidini r days | |
| MGMT | | | X |
| methylation status | | | ^ |
| (see Section 4 for | | | |
| details) | | | |
| Tissue, blood, | | | X |
| urine for banking | | | |
| (if patient | | | |
| consents; see | | | |
| Section 10 for | | | |
| details) | | | |

**Assessments During Treatment** 

| | ASSESSITIET | its During Treatment |
|---|---|---|
| Assessment | q8 weeks (± 3 days) | At 8 weeks, 24 weeks, and progression |
| Physical | RT arm: weekly during RT | |
| | Non-RT arm: q8 weeks | |
| Weight | X (See 7.1.1; done prior to | |
| | each drug dose) | |
| Neurological exam | X | |
| Tumor imaging | X | |
| MRI/CT scan | | |
| Karnofsky status | X | |
| CBC w/ differential | X | |
| Urine protein: | X (See 11.1; done prior to | |
| creatinine or urine | each drug dose) | |
| dipstick | | |
| MR diffusion and | | X |
| perfusion imaging | | |
| (optional but strongly | | |
| recommended) | | |
| Blood pressure | X (See 11.1; done prior to | |
| monitoring | each drug dose) | |
| AE evaluation | X | |
| Blood, urine for | At 8 weeks after treatment | |
| banking | initiation (± 3 days) | |
| (if patient consents) | | |

Follow-Up Assessments

| Assessments | After treatment discontinuation or progression: q8 weeks for 1 year, then q6 months for 1 year, then annually (± 2 weeks). (See Section 12.1 for details) |
|---|---|
| Physical | X |
| Karnofsky status | X |
| AE evaluation | X |

#### **APPENDIX II**

### KARNOFSKY PERFORMANCE SCALE

| 100 | Normal; no complaints; no evidence of disease |
|-----|-----------------------------------------------------------------------|
| 90 | Able to carry on normal activity; minor signs or symptoms of disease |
| 80 | Normal activity with effort; some sign or symptoms of disease |
| 70 | Cares for self; unable to carry on normal activity or do active work |
| 60 | Requires occasional assistance, but is able to care for most personal |
| | needs |
| 50 | Requires considerable assistance and frequent medical care |
| 40 | Disabled; requires special care and assistance |
| 30 | Severely disabled; hospitalization is indicated, although death not |
| | imminent |
| 20 | Very sick; hospitalization necessary; active support treatment is |
| | necessary |
| 10 | Moribund; fatal processes progressing rapidly |
| 0 | Dead |

#### **APPENDIX III** (10/9/14)

Appendices for NRG Oncology Biospecimen Collection (as specified by the protocol).

NRG Oncology FFPE Specimen Plug Kit Collection NRG Oncology Blood Collection Kit Instructions NRG Oncology Urine Collection Kit Instructions

#### **Shipping Instructions:**

U.S. Postal Service Mailing Address: <u>For FFPE or Non-frozen Specimens Only</u> NRG Oncology Biospecimen Bank
University of California San Francisco
UCSF Box 1800
2340 Sutter Street, Room S341
San Francisco, CA 94143-1800

Courier Address (FedEx, UPS, etc.): <u>For Frozen or Trackable Specimens</u> NRG Oncology Biospecimen Bank University of California San Francisco 2340 Sutter Street, Room S341 San Francisco, CA 94115

- □ Include all NRG Oncology paperwork in pocket of biohazard bag.
- □ Check that the Specimen Transmittal (ST) Form has the consent boxes checked off.
- □ Check that all samples are labeled with the NRG Oncology study and case number, and include date of collection as well as collection time point (e.g., pretreatment, post-treatment).

#### □ FFPE Specimens:

- Slides should be shipped in a plastic slide holder/slide box. Place a small wad of padding in top
  of the container. If you can hear the slides shaking it is likely that they will break during
  shipping.
- FFPE Blocks can be wrapped in paper or placed in a cardboard box with padding. Do not wrap blocks with bubble wrap or gauze. Place padding in top of container so that if you shake the container the blocks are not shaking If you can hear the block shaking it might break during shipping.
- Slides, Blocks, or Plugs can be shipped ambient or with a cold pack either by United States Postal Service (USPS) to the USPS address (94143) or by Courier to the Street Address (94115). Do NOT ship on Dry Ice.

#### □ Frozen Specimens:

- Multiple cases may be shipped in the same cooler, but make sure each one is in a separate bag and clearly identified. . If possible keep Serum, Plasma, and Whole Bloods in separate bags.
- Place specimens and absorbent shipping material in Styrofoam cooler filled with dry ice (at least 7 lbs). There should be plenty of dry ice under and above the specimens. If the volume of specimens is greater than the volume of dry ice then ship in a larger Styrofoam box, or two separate boxes. Any Styrofoam box can be used, as long as it is big enough.
- Specimens received thawed due to insufficient dry ice or shipping delays will be discarded and the site will be notified.
- Send frozen specimens on dry ice via overnight courier to the address above. Specimens should only be shipped Monday through Wednesday (Monday-Tuesday for Canada) to prevent thawing due to delivery delays. Saturday or holiday deliveries cannot be accepted. Samples can be stored frozen at -80° C until ready to ship.
- □ For Questions regarding collection/shipping please contact the NRG Oncology Biospecimen Bank by e-mail: <a href="mailto:RTOG@ucsf.edu">RTOG@ucsf.edu</a> or phone: 415-476-7864 or Fax: 415-476-5271.

#### NRG ONCOLOGY FFPE SPECIMEN PLUG KIT INSTRUCTIONS

This Kit allows sub-sampling of an FFPE block for submission to the NRG Oncology Biospecimen Bank. The plug kit contains a shipping tube and a punch tool.



#### Step 1

If the block is stored cold, allow it to equilibrate for 30 minutes at room temperature. Place the punch tool on the paraffin block over the selected tumor area. (Ask a pathologist to select area with tumor.) Push the punch into the paraffin block. Twist the punch tool once around to separate the plug from the block. Then pull the punch tool out of the block. The punch should be filled with tissue sample.



#### Step 2

Label the punch tool with the proper specimen ID. Include the pathology accession number and block ID. DON'T remove specimen from the punch.

Use a separate punch tool for every specimen. Call or e-mail us if you have any questions or need additional specimen plug kits.



#### Step 3

Once punch tool is labeled, place in shipping tube and mail to address below. Please do not mix specimens in the same tube.

We will remove core specimen from the punch, embed in a paraffin block, and label with specimen ID.

\*NOTE: If your facility is uncomfortable obtaining the plug but wants to retain the tissue block, please send the entire block to the NRG Oncology Biospecimen Bank and we will sample a plug from the block and return the remaining block to your facility. Please indicate on the submission form the request to perform the plug procedure and return of the block.

Ship specimen plug kit, specimen in punch tool, and all paperwork to the address below. For Questions regarding collection/shipping or to order an FFPE Specimen Plug Kit, please contact the NRG Oncology Biospecimen Bank by e-mail: RTOG@ucsf.edu or call 415-476-7864/Fax 415-476-5271.

| U.S. Postal Service Mailing Address: | Courier Address (FedEx, UPS, etc.): |
|---|---|
| For Non-frozen Specimens Only | For Frozen Specimens or Trackable |
| | shipments |
| NRG Oncology Biospecimen Bank | |
| University of California San Francisco | NRG Oncology Biospecimen Bank |
| UCSF Box 1800 | University of California San Francisco |
| 2340 Sutter Street, Room S341 | 2340 Sutter Street, Room S341 |
| San Francisco, CA 94143-1800 | San Francisco, CA 94115 |

#### NRG ONCOLOGY BLOOD COLLECTION KIT INSTRUCTIONS

This Kit is for collection, processing, storage, and shipping of <u>serum</u>, <u>plasma</u>, <u>or whole blood</u> (as specified by the protocol):

#### Kit contents:

- One Red Top tube for serum (A)
- One Purple Top EDTA tube for plasma (B)
- One Purple Top EDTA tube for Whole Blood (C)
- Twenty-one (21) 1 ml cryovials
- Biohazard bags (3) and Absorbent shipping material (3)
- Styrofoam container (inner) and Cardboard shipping (outer) box
- UN1845 DRY Ice Sticker and UN3373 Biological Substance Category B Stickers
- Specimen Transmittal (ST) Form and Kit Instructions

#### PREPARATION AND PROCESSING OF SERUM, PLASMA AND WHOLE BLOOD:

#### (A) Serum (if requested): Red Top Tube

□ Label as many 1ml cryovials (5 to 8) as necessary for the serum collected. Label them with the NRG Oncology study and case number, collection date, time, and time point, and clearly mark cryovials "serum".

#### Process:

- 1. Allow one red top tube to clot for 30 minutes at room temperature.
- 2. Spin in a standard clinical centrifuge at ~2500 RPM for 10 minutes at 4°C (preferred). If sites are unable to process samples at 4°C then spinning at room temperature is acceptable if done within 2 hours of draw but must be noted on the ST Form.
- 3. Aliquot 0.5 ml serum into as many cryovials as are necessary for the serum collected (5 to 8) labeled with NRG Oncology study and case numbers, collection date/time, protocol time-point collected (e.g. pretreatment, post-treatment), and clearly mark specimen as "serum". If an aliquot has less than 0.5 ml in the tube please note the volume on the vial and make a note on the ST Form.
- 4. Place cryovials into biohazard bag and immediately freeze at -70 to -90° C, and store frozen until ready to ship. See below for storage conditions.
- 5. Store serum at -70 to -90° C until ready to ship on dry ice. See below for storage conditions.

## PLEASE MAKE SURE THAT EVERY SPECIMEN IS LABELED and include collection time point on the ST Form.

#### (B) Plasma (If requested): Purple Top EDTA tube #1

□ Label as many 1ml cryovials (5 to 8) as necessary for the plasma collected. Label them with the NRG Oncology study and case number, collection date, time, and time point, and clearly mark cryovials "plasma".

#### **Process:**

- 1. After collection, invert tube(s) multiple times to ensure adequate mixing of EDTA.
- 2. Centrifuge specimen(s) within one hour of collection in a standard clinical centrifuge at ~2500 RPM for 10 minutes at 4°C (preferred). If sites are unable to process samples at 4°C then spinning at room temperature is acceptable if done within 2 hours of draw but must be noted on the ST Form.
- 3. If the interval between specimen collection and processing is anticipated to be more than one hour, keep specimen on ice until centrifuging is performed.
- 4. Carefully pipette and aliquot 0.5 ml plasma into as many cryovials as are necessary for the plasma collected (5 to 8) labeled with NRG Oncology study and case numbers, collection date/time, time point collected and clearly mark specimen as "plasma". Avoid pipetting up the buffy coat layer. If an aliquot has less than 0.5 ml in the tube please note the volume on the vial and make a note on the ST Form.
- 5. Place cryovials into biohazard bag and immediately freeze at -70 to -90°C.
- 6. Store frozen plasma until ready to ship on dry ice.
- 7. See below for storage conditions.

## PLEASE MAKE SURE THAT EVERY SPECIMEN IS LABELED and include collection time point on the ST Form.



#### (C) Whole Blood for DNA (if requested): Purple Top EDTA tube #2

□ Label as many 1ml cryovials (3 to 5) as necessary for the whole blood collected. Label them with the NRG Oncology study and case number, collection date/time, and time point, and clearly mark cryovials "blood".

#### **Process:**

- 1. After collection, invert tube(s) multiple times to ensure adequate mixing of EDTA. Blood can also be mixed for 5 minutes on a mixer at room temperature.
- Carefully pipette and aliquot 1.0 ml blood into as many cryovials as are necessary for the blood collected (3 to 5) labeled with NRG Oncology study and case numbers, collection date/time, time point collected and clearly mark specimen as "blood". If an aliquot has less than 1.0 ml in the tube please note the volume on the vial and make a note on the ST Form.
- 3. Place cryovials into biohazard bag and freeze immediately at -70 to -80° Celsius.
- 4. Store blood samples frozen until ready to ship on dry ice.
- 5. See below for storage conditions.

## PLEASE MAKE SURE THAT EVERY SPECIMEN IS LABELED and include collection time point on ST Form.

#### Freezing and Storage:

- ☐ Freeze Blood samples in a -80°C Freezer or on Dry Ice or snap freeze in liquid nitrogen.
- □ Store at −80°C (-70°C to -90°C) until ready to ship.
  - If a -80°C Freezer is not available,
    - Samples can be stored short term in a -20°C freezer (non-frost free preferred) for up to one week (please ship out Monday-Wednesday only; Canada: Monday-Tuesday only).

#### OR:

Samples can be stored in plenty of dry ice for up to one week, replenishing daily (please ship out on Monday-Wednesday only; Canada: Monday-Tuesday only).

#### OR:

- Samples can be stored in liquid nitrogen vapor phase (ship out Monday-Wednesday only; Canada: Monday-Tuesday only).
- Please indicate on Specimen Transmittal Form the storage conditions used and time stored.

#### Shipping/Mailing:

□ Ship specimens on Dry Ice overnight **Monday-Wednesday (Monday-Tuesday from Canada)** to prevent thawing due to delivery delays. Saturday and holiday deliveries cannot be accepted.

- Include all NRG Oncology paperwork in a sealed plastic bag and tape to the outside top of the Styrofoam box.
- □ Wrap frozen specimens of same type (i.e., all serum together, plasma together and whole bloods together) in absorbent shipping material and place each specimen type in a separate biohazard bag. Place specimen bags into the Styrofoam cooler and fill with plenty of dry ice (7-10 lbs/3.5kg minimum). Add padding to avoid the dry ice from breaking the tubes.
- □ Place Styrofoam coolers into outer cardboard box, and attach shipping label and UN3373 and UN1895 stickers to outer cardboard box.
- Multiple cases may be shipped in the same cooler, but make sure each one is in a separate bag and that there is enough room for plenty of dry ice. Add padding to avoid the dry ice from breaking the tubes.
- □ For questions regarding collection, shipping or to order a Blood Collection Kit, please e-mail RTOG@ucsf.edu or call (415)476-7864.

#### **Shipping Address:**

Courier Address (FedEx, UPS, etc.): For all Frozen Specimens NRG Oncology Biospecimen Bank San Francisco University of California San Francisco 2340 Sutter Street, Room S341 San Francisco, CA 94115 For questions, call 415-476-7864 or e-mail: RTOG@ucsf.edu

#### NRG ONCOLOGY URINE COLLECTION KIT INSTRUCTIONS

This Kit is for collection, processing, storage, and shipping of urine specimens. Kit Contents:

- One (1) Sterile Urine collection cup
- Two 7 ml disposable pipettes
- Absorbent paper towel

- Two 15 ml polypropylene centrifuge tubes
- Biohazard bags
- Parafilm for sealing outside of tubes

#### **Preparation and Processing of Urine Specimens:**

#### Process:

- A clean catch urine specimen will be collected. To collect the specimen, use the following instructions:
  - Males should wipe clean the head of the penis and females need to wipe between the labia with soapy water/cleansing wipes to remove any contaminants.
  - After urinating a small amount into the toilet bowl to clear the urethra of contaminants, collect a sample of urine in the collection cup.
  - After 10-25 mL urine has been collected, remove the container from the urine stream without stopping the flow of urine.
  - Finish voiding the bladder into the toilet bowl.
- Aliquot 5-10 mls of Urine into each of two 15 ml polypropylene centrifuge tubes (disposable
  pipets are provided in the kit). Do not fill with more than 10 mls to avoid cracking of tubes due
  to expansion during freezing. Replace the cap and tighten on the tubes. Make sure the cap is
  not cross-threaded or placed on incorrectly or leaking will occur.
- Use parafilm to seal the cap around the outside rim of the urine tube to prevent leakage.
- Discard remaining Urine and collection cup.
- Label the specimen with the NRG Oncology study and case number, collection date and time, time point of collection, and clearly mark specimens as "urine".
- Wrap Urine Tubes with absorbent material (paper towels) and place into biohazard bag and seal the bag. Freeze and store Urine samples in a -20°C or -80°C freezer until ready to ship.

PLEASE MAKE SURE THAT EVERY SPECIMEN IS LABELED with NRG Oncology study and case numbers, collection date/time, and time point collected (e.g. pretreatment, post-treatment).

#### **Storage and Shipping:**

#### Freezing and Storage:

- □ Urine specimens may be sent in batches or with other frozen biospecimens, if within 30-60 days of collection. Store at -20°C or -80°C (-70°C to -90°C) until ready to ship. If a -80°C Freezer is not available:
  - Samples can be stored short term in a -20° C freezer (non-frost free preferred) for up to one week (please ship out Monday-Wednesday only; Canada: Monday-Tuesday only).

#### OR:

- Samples can be stored in plenty of Dry Ice for up to one week, replenishing daily (please ship out Monday-Wednesday only; Canada: Monday-Tuesday only).
- Please indicate on Specimen Transmittal Form the storage conditions used and time stored.

#### Shipping/Mailing:

- Ship specimens on Dry Ice overnight **Monday-Wednesday (Monday-Tuesday from Canada)** to prevent thawing due to delivery delays. Saturday and holiday deliveries cannot be accepted.
- ☐ Include all NRG Oncology paperwork in a sealed plastic bag and tape to the outside top of the Styrofoam box.
- □ Place sealed specimen bags into the Styrofoam cooler and fill with plenty of dry ice (7-10 lbs/3.5kg minimum). *Add padding to avoid the dry ice from breaking the tubes.*
- Place Styrofoam coolers into outer cardboard box, and attach shipping label and UN3373 and UN1895 stickers to outer cardboard box.

- Multiple cases may be shipped in the same cooler, but make sure each one is in a separate bag and that there is enough room for plenty of dry ice. Add padding to avoid the dry ice from breaking the tubes.
- □ Samples received thawed will be discarded, and a notification will be sent immediately to the Principal Investigator and Clinical Research Assistant of the submitting institution. The institution should send a subsequent sample, collected as close as possible to the original planned collection date.
- □ For questions regarding ordering, collection, or shipping of a Urine Collection Kit, please e-mail RTOG@ucsf.edu or call (415)476-7864 or fax (415) 476-5271.

Shipping Address: FedEx/UPS/Courier address (For all frozen samples)
NRG Oncology Biospecimen Bank San Francisco
2340 Sutter Street, Room S341, UCSF
San Francisco, CA 94115
Contact Phone: (415) 476-7864